CLINICAL TRIAL: NCT00521586
Title: A Phase 3, Randomized, Double-blind Trial To Evaluate The Safety, Tolerability, And Immunogenicity Of A 13-valent Pneumococcal Conjugate Vaccine (13vpnc) When Administered Concomitantly With Trivalent Inactivated Influenza Vaccine In Healthy Adults 50-59 Years Of Age Who Are Naive To 23-valent Pneumococcal Polysaccharide Vaccine And To Evaluate The Immune Response Of A Second Dose Of 13vpnc Administered 5 Years After Initial 13vpnc Vaccination
Brief Title: Study Evaluating 13 Valent Pneumococcal Conjugate Vaccine With Trivalent Inactivated Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 6115A1-3001; B1851020 (Other: Alias Study Number)
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Influenza
Keywords: Pneumococcal Conjugate Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): arm 1 = TIV +13vPnC at visit 1, placebo at visit 2 then 13vPnC at year 5
  Interventions: Biological: 13 valent pneumococcal conjugate vaccine
- 2 (Other): arm 2 = TIV + placebo at visit 1, then 13vPnC at visit 2 and at year 5
  Interventions: Biological: 13 valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13 valent pneumococcal conjugate vaccine — TIV +13vPnC at dose 1 placebo at dose 2, one month after dose 1 13vPnC at year 5
  Other Names: 0.5 mL dose of TIV and 13vPnC at dose 1, 0.5 mL dose of of placebo at dose 2, and 0.5ml dose of 13vPnC at year 5 will be administered into left deltoid muscle
  Arms: 1
Biological: 13 valent pneumococcal conjugate vaccine — TIV + placebo at dose 1 13vPnC at dose 2, one month after dose 1 and 13vPnC at year 5
  Other Names: 0.5 mL dose of TIV and of placebo at dose 1 and 0.5 mL dose of 13vPnC at dose 2 and year 5 will be administered into left deltoid muscle
  Arms: 2

SUMMARY:
This study is to evaluate the safety, tolerability and immune response when 13-valent pneumococcal conjugate vaccine (13vPnC) and the trivalent inactivated flu vaccine (TIV) are given together to healthy adults aged 50-59 years who are naive to 23-valent pneumococcal polysaccharide vaccine (23vPS), or when the vaccines are given 1 month apart. It will also evaluate the immune response to 13vPnC once per year for 4 years and then to a second dose of 13vPnC given 5 years after the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 50 to 59 years
* Determined by medical history, physical examination and clinical judgement to be eligible for the study
* Able to complete electronic diary
* Available for the 5 year 9 month duration of the study

Exclusion Criteria:

* Previous vaccination with any licensed or experimental pneumococcal vaccine
* Allergic to egg proteins and chicken proteins
* History of Guillian-Barre syndrome
* Vaccination with TIV within 6 months before study start
* Vaccination with diphtheria-containing vaccine within 6 months of study start
* Serious chronic disorders including immunodeficiency or metastatic malignancy
* Known or suspected hypersensitivity to any vaccine or vaccine component

Ages: 50 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1116 (Actual)
Dates: Start 2007-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (39):
  - Clinical Research Advantage, Inc., Chandler, Arizona
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Clinical Trials Center Pediatric Infectious Diseases and Clinical Trials, Aurora, Colorado
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - A. G. A. Clinical Trials, Hialeah, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Accelovance, Peoria, Illinois
  - Suite 100, Riverdale, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Radiant Research, Inc, St Louis, Missouri
  - Big Sky Clinical Research, Butte, Montana
  - FFM Clinical Research, Camillus, New York
  - Rochester Clinical Research, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - PMG Research of Raleigh, LLC, Cary, North Carolina
  - Hickory Family Practice Associates, Hickory, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Unifour Medical Research Associates, LLC, Hickory, North Carolina
  - Unifour Medical Research Associates, Hickory, North Carolina
  - Fairbrook Medical Clinic, Hickory, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center Gamble Program for Clinical Studies, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Preferred Primary Care Physicians, Inc, Carnegie, Pennsylvania
  - Family Healthcare Partners, Grove City, Pennsylvania
  - Family Practice Medical Associates South, Jefferson Office, Jefferson Hills, Pennsylvania
  - Kid's Plus Pediatrics, Pittsburgh, Pennsylvania
  - Primary Physicians Research Inc., Pittsburgh, Pennsylvania
  - Family Practice Medical Associates South, Upper Saint Clair, Pennsylvania
  - The Washington Hospital Family Medicine, Washington, Pennsylvania
  - Internal Medicine & Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Clark D. McKeever, M.D. Research for Health, Houston, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Advanced Clinical Research, West Jordan, Utah

REFERENCES:
- [Derived] Frenck RW Jr, Fiquet A, Gurtman A, van Cleeff M, Davis M, Rubino J, Smith W, Sundaraiyer V, Sidhu M, Emini EA, Gruber WC, Scott DA, Schmoele-Thoma B; B1851020 Study Group. Immunogenicity and safety of a second administration of 13-valent pneumococcal conjugate vaccine 5 years after initial vaccination in adults 50 years and older. Vaccine. 2016 Jun 24;34(30):3454-62. doi: 10.1016/j.vaccine.2016.04.093. Epub 2016 May 5. PMID 27155493
- [Derived] Frenck RW Jr, Gurtman A, Rubino J, Smith W, van Cleeff M, Jayawardene D, Giardina PC, Emini EA, Gruber WC, Scott DA, Schmole-Thoma B. Randomized, controlled trial of a 13-valent pneumococcal conjugate vaccine administered concomitantly with an influenza vaccine in healthy adults. Clin Vaccine Immunol. 2012 Aug;19(8):1296-303. doi: 10.1128/CVI.00176-12. Epub 2012 Jun 27. PMID 22739693
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-3001&StudyName=Study%20Evaluating%20%2013%20Valent%20Pneumococcal%20Conjugate%20Vaccine%20with%20Trivalent%20Inactivated%20Influenza%20Vaccine

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initially 1060 participants were reported to complete the 6 month follow up at Year 0, however 6 additional participants who were reported to have withdrawn initially, actually completed the 6 month follow up at Year 0.
Groups:
- 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5): Participants received 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscular injection into the deltoid muscle of the left arm along with 0.5-mL trivalent inactivated influenza vaccine (TIV) intramuscular injection into the deltoid muscle of the right arm at Year 0 on Day 1 (Dose 1, 13vPnC+TIV). Placebo matched to 13vPnC was administered 1 month after (Dose 2, placebo). Participants were further followed-up for 1 month, then attended a 6-month follow-up visit for safety. Participants were then followed-up yearly for 4 years. Participants then received 0.5 mL dose of 13vPnC intramuscular injection into the deltoid muscle of the left arm 5 years after initial vaccination. Participants were further followed-up for 1 month, then attended a 6-month follow-up visit for safety.
- Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5): Participants received placebo matched to 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscular injection into the deltoid muscle of the left arm along with 0.5-mL trivalent inactivated influenza vaccine (TIV) intramuscular injection into the deltoid muscle of the right arm at Year 0 on Day 1 (Dose 1, placebo+TIV). 13vPnC was administered 1 month after (Dose 2, 13vPnC). Participants were further followed-up for 1 month, then attended a 6-month follow-up visit for safety. Participants were then followed-up yearly for 4 years. Participants then received 0.5 mL dose of 13vPnC intramuscular injection into the deltoid muscle of the left arm 5 years after initial vaccination. Participants were further followed-up for 1 month, then attended a 6-month follow-up visit for safety.
Period: Initial Vaccination (Year 0)
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Started | 554 | 562
Vaccinated Dose 1 | 551 | 560
Vaccinated Dose 2 | 538 | 543
Initially Reported to Complete Year 0 | 531 (Initially 1060 participants were reported to complete follow-up(Year 0),but 1066 actually completed.) | 529 (Initially 1060 participants were reported to complete follow-up(Year 0),but 1066 actually completed.)
Completed | 533 (6 additional participants initially reported to have withdrawn, actually completed follow-up(Year 0)) | 533 (6 additional participants initially reported to have withdrawn, actually completed follow-up(Year 0))
Not Completed | 21 | 29
Not completed — Subject request | 8 | 11
Not completed — Lost to Follow-up | 5 | 10
Not completed — Protocol Violation | 2 | 5
Not completed — Other, unspecified | 3 | 1
Not completed — Investigator request | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 0
Not completed — Failed to return | 0 | 1
Period: Follow-up (From 6-month[Year 0]-Year 5)
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Started | 533 | 533
Completed | 364 | 363
Not Completed | 169 | 170
Not completed — Adverse Event | 5 | 1
Not completed — Death | 5 | 2
Not completed — Failed to return | 7 | 3
Not completed — Investigator request | 3 | 3
Not completed — Lost to Follow-up | 55 | 56
Not completed — Other | 22 | 26
Not completed — Protocol Violation | 18 | 22
Not completed — Subject request | 54 | 57
Period: Revaccination With 13vPnC (Year 5)
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Started | 364 | 363
Vaccinated 13vPnC (Year 5) | 364 | 363
Completed 1 Month Follow-up | 363 | 359
Completed 6 Month Follow-up | 361 | 351
Completed | 361 | 351
Not Completed | 3 | 12
Not completed — Subject request | 0 | 1
Not completed — Failed to return | 1 | 4
Not completed — Lost to Follow-up | 2 | 7

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who had received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5) | Total
Number analyzed (Participants) | 551 | 560 | 1111
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (2.8) | 54.6 (2.9) | 54.6 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 319 | 322 | 641
  Male | 232 | 238 | 470

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving at Least 4-fold Increase in Titer for Concomitant Trivalent Inactivated Influenza Vaccine (TIV) Antigens 1 Month After Dose 1
Description: Percentage of participants achieving at least 4-fold increase in titer for concomitant Trivalent Inactivated Influenza Vaccine (TIV) were measured by standard Hemagglutination Inhibition Assay (HAI) for the A/H1, A/H3, and B vaccine strains.Exact, unconditional, 2-sided, 95% confidence intervals (CI) on the difference in proportions (13vPnC+TIV - Placebo+TIV) was calculated. N(number of participants analyzed)=participants with a determinate antibody titer to the given concomitant vaccine antigen. n=participants who met the prespecified level for the given antigen.
Time Frame: 1 month after Dose 1
Population: Evaluable immunogenicity population:eligible participants who received vaccination as assigned;had blood drawn within pre-specified time-frames;had at least 1 valid,determinate assay result;had no major protocol violation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 530 | 531
percentage of participants
  A/H1N1 strain (n=445,431) | 84.0 [80.6 to 87.0] | 81.2 [77.6 to 84.4]
  A/H3N2 strain (n=377,369) | 71.1 [67.1 to 75.0] | 69.5 [65.4 to 73.4]
  B strain (n=321,320) | 60.6 [56.3 to 64.8] | 60.3 [56.0 to 64.5]
Statistical Analysis 1: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); A/H1N1 strain: Exact 2-sided, 95 percent (%) confidence intervals was computed based on the methodology by Chan and Zhang; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower limit of the 2-sided 95% CI was greater than -0.1 or -10%; percent difference = 2.8, 95% CI 2-sided [-1.8 to 7.4]
Statistical Analysis 2: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); A/H3N2 strain: Exact 2-sided, 95 % confidence intervals was computed based on the methodology by Chan and Zhang; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower limit of the 2-sided 95% CI was greater than -0.1 or -10%; percent difference = 1.6, 95% CI 2-sided [-3.9 to 7.2]
Statistical Analysis 3: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); B strain: Exact 2-sided, 95 % confidence intervals was computed based on the methodology by Chan and Zhang; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower limit of the 2-sided 95% CI was greater than -0.1 or -10%; percent difference = 0.3, 95% CI 2-sided [-5.6 to 6.2]

2. Primary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After 13vPnC Dose
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) for adult participants are presented. GMC (13vPnC) and corresponding 2-sided 95 percent (%) CIs were evaluated. Geometric means were calculated using all participants with available data for 1 month after 13vPnC Dose at year 0 blood draw. CI for GMC are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: 1 month after 13vPnC Dose at year 0
Population: Evaluable immunogenicity population:eligible participants who received vaccination as assigned;had blood drawn within pre-specified time-frames;had at least 1 valid,determinate assay result;had no major protocol violation. n=participants with valid and determinate assay results for the specified serotype at the given visit.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 531 | 532
microgram per milliliter (mcg/mL)
  Serotype 1 (n=292, 289) | 4.05 [3.41 to 4.81] | 5.45 [4.57 to 6.49]
  Serotype 3 (n=290, 288) | 1.15 [1.02 to 1.29] | 1.46 [1.29 to 1.65]
  Serotype 4 (n=290, 288) | 2.35 [2.00 to 2.77] | 3.41 [2.89 to 4.02]
  Serotype 5 (n=293, 289) | 6.03 [5.16 to 7.05] | 7.18 [6.13 to 8.40]
  Serotype 6A (n=293, 288) | 5.78 [5.02 to 6.64] | 6.70 [5.74 to 7.83]
  Serotype 6B (n=292, 289) | 7.58 [6.54 to 8.78] | 10.09 [8.57 to 11.86]
  Serotype 7F (n=293, 289) | 8.14 [7.07 to 9.38] | 10.57 [9.11 to 12.27]
  Serotype 9V (n=293, 289) | 4.96 [4.32 to 5.70] | 6.97 [6.08 to 7.99]
  Serotype 14 (n=294, 288) | 10.77 [9.04 to 12.82] | 14.05 [11.82 to 16.71]
  Serotype 18C (n=293, 288) | 9.65 [8.32 to 11.19] | 13.49 [11.62 to 15.67]
  Serotype 19A (n=294, 289) | 16.80 [14.75 to 19.14] | 18.84 [16.37 to 21.68]
  Serotype 19F (n=291, 286) | 6.13 [5.21 to 7.22] | 7.13 [5.90 to 8.63]
  Serotype 23F (n=294, 289) | 7.17 [6.06 to 8.49] | 8.54 [7.11 to 10.25]
Statistical Analysis 1: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 1: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — Noninferiority was to be concluded if the lower limit of the 2-sided 95% CI for the GMR was greater than 0.5 (2-fold criterion); Geometric mean ratio = 0.74, 95% CI 2-sided [0.58 to 0.95]
Statistical Analysis 2: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 3: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.79, 95% CI 2-sided [0.66 to 0.93]
Statistical Analysis 3: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 4: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.69, 95% CI 2-sided [0.55 to 0.87]
Statistical Analysis 4: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 5: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.84, 95% CI 2-sided [0.67 to 1.05]
Statistical Analysis 5: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 6A: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.86, 95% CI 2-sided [0.70 to 1.06]
Statistical Analysis 6: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 6B: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.75, 95% CI 2-sided [0.60 to 0.93]
Statistical Analysis 7: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 7F: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.77, 95% CI 2-sided [0.63 to 0.95]
Statistical Analysis 8: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 9V: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.71, 95% CI 2-sided [0.59 to 0.86]
Statistical Analysis 9: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 14: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.60 to 0.98]
Statistical Analysis 10: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 18C: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 0.72, 95% CI 2-sided [0.58 to 0.88]
Statistical Analysis 11: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 19A: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 0.89, 95% CI 2-sided [0.74 to 1.08]
Statistical Analysis 12: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 19F: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 0.86, 95% CI 2-sided [0.67 to 1.10]
Statistical Analysis 13: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); Serotype 23F: 2-sided 95 % CI for the ratio of 2 geometric means (13vPnC+TIV/Placebo and Placebo+TIV/13vPnC) was constructed by back transformation of the CIs for the difference of the 2 logarithmically transformed assay results computed using the Student t distribution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 0.84, 95% CI 2-sided [0.66 to 1.08]

3. Other Pre Specified Outcome: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT) 1 Month After 13vPnC (Year 5)
Description: Serotype-specific OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of participants using a microcolony OPA (mcOPA) assay. GMTs (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data for 1 Month After 13vPnC (Year 5) blood draws. CI for GMTs were back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 1 month after 13vPnC (Year 5)
Population: All-available immunogenicity population at Year 5 included participants who had at least 1 valid and determinate assay result related to the proposed analysis. n=participants with valid and determinate assay results for the specified serotype at 1 month after 13vPnC (Year 5) blood draws for each treatment arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5): Participants received 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscular injection into the deltoid muscle of the left arm along with 0.5-mL trivalent inactivated influenza vaccine (TIV) intramuscular injection into the deltoid muscle of the right arm on Day 1(Dose 1). Placebo matched to 13vPnC vaccine (dose 2) was administered 1 month after vaccination 1, dose 1 (13vPnC+TIV).Participants were then followed-up to 4 years (for 1 month, then 6 month and then yearly follow-up) after dose 2 of vaccination 1. Participants then received 0.5 mL dose of 13vPnC vaccine intramuscular injection into the deltoid muscle of the left arm 5 years after vaccination 1. Participants were further followed-up for 1 month and then for 6 months.
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 363 | 363
titers
  Serotype 1 (n=349,352 ) | 178 [150.6 to 210.1] | 168 [141.4 to 199.9]
  Serotype 3(n=355, 352) | 59 [52.1 to 67.1] | 66 [57.7 to 75.0]
  Serotype 4(n=357,350) | 1618 [1453.2 to 1801.5] | 1491 [1318.4 to 1685.8]
  Serotype 5(n=350,353) | 267 [224.7 to 317.0] | 312 [266.2 to 366.6]
  Serotype 6A(n=356,350) | 4266 [3752.0 to 4849.9] | 3994 [3442.0 to 4635.6]
  Serotype 6B(n=354,351) | 3583 [3130.7 to 4101.8] | 3567 [3149.2 to 4040.9]
  Serotype 7F(n=355,352) | 1636 [1459.8 to 1834.3] | 1803 [1624.6 to 2001.7]
  Serotype 9V(n=353,347) | 1818 [1581.5 to 2090.6] | 1551 [1282.4 to 1875.8]
  Serotype 14(n=355,350) | 1110 [993.2 to 1239.7] | 1107 [988.1 to 1240.1]
  Serotype 18C(n=353,348) | 1800 [1571.8 to 2060.7] | 1738 [1485.4 to 2033.8]
  Serotype 19A(n=354,352) | 913 [815.7 to 1022.9] | 890 [787.1 to 1006.5]
  Serotype 19F(n=345,338) | 1202 [1030.9 to 1402.0] | 1140 [976.7 to 1330.3]
  Serotype 23F(n=354,350) | 1837 [1562.6 to 2159.9] | 1820 [1552.0 to 2134.4]
Statistical Analysis 1: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Geometric Mean Ratio = 1.1, 95% CI 2-sided [0.83 to 1.34]
Statistical Analysis 2: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; Geometric Mean Ratio = 0.9, 95% CI 2-sided [0.75 to 1.08]
Statistical Analysis 3: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; Geometric Mean Ratio = 1.1, 95% CI 2-sided [0.92 to 1.28]
Statistical Analysis 4: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; Geometric Mean Ratio = 0.9, 95% CI 2-sided [0.68 to 1.08]
Statistical Analysis 5: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; Geometric Mean Ratio = 1.1, 95% CI 2-sided [0.88 to 1.30]
Statistical Analysis 6: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; Geometric Mean Ratio = 1.0, 95% CI 2-sided [0.84 to 1.21]
Statistical Analysis 7: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; Geometric Mean Ratio = 0.9, 95% CI 2-sided [0.78 to 1.06]
Statistical Analysis 8: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; Geometric Mean Ratio = 1.2, 95% CI 2-sided [0.93 to 1.48]
Statistical Analysis 9: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; Geometric Mean Ratio = 1.0, 95% CI 2-sided [0.86 to 1.17]
Statistical Analysis 10: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; Geometric Mean Ratio = 1.0, 95% CI 2-sided [0.84 to 1.27]
Statistical Analysis 11: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; Geometric Mean Ratio = 1.0, 95% CI 2-sided [0.87 to 1.21]
Statistical Analysis 12: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 12]; Test type: Superiority or Other; Geometric Mean Ratio = 1.1, 95% CI 2-sided [0.85 to 1.31]
Statistical Analysis 13: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; Geometric Mean Ratio = 1.0, 95% CI 2-sided [0.80 to 1.27]

4. Other Pre Specified Outcome: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) Before 13vPnC (Year 5) and 1 Month After 13vPnC Re-vaccinated Dose (Year 5)
Description: Serotype-specific OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of participants using a microcolony OPA (mcOPA) assay. GMTs (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data for before 13vPnC (Year 5) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws. CI for GMTs were back transformations of a CI based on the Student t distribution for the mean logarithm of the titers. Participants with immunogenicity data at both Year 5 endpoints.
Time Frame: before 13vPnC (Year 5) and 1 month after 13vPnC re-vaccinated dose (Year 5)
Population: All-available immunogenicity population at Year 5.n=participants with valid and determinate assay results for the specified serotype at before 13vPnC (Year 5) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws for each treatment arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- All Participants: Participants received either 0.5 mL dose of 13vPnC intramuscular injection into the deltoid muscle of the left arm along with 0.5-mL TIV intramuscular injection into the deltoid muscle of the right arm at Year 0 on Day 1 (Dose 1, 13vPnC+TIV), or placebo matched to 13vPnC intramuscular injection into the deltoid muscle of the left arm along with 0.5-mL TIV intramuscular injection into the deltoid muscle of the right arm at Year 0 on Day 1 (Dose 1, placebo+TIV). One month after, participants received either Placebo matched to 13vPnC (Dose 2, placebo), or 13vPnC (Dose 2, 13vPnC). Participants were further followed-up for 1 month, then attended a 6-month follow-up visit for safety. Participants were then followed-up yearly for 4 years. Participants then received 0.5 mL dose of 13vPnC intramuscular injection into the deltoid muscle of the left arm 5 years after initial vaccination. Participants were further followed-up for 1 month, then attended a 6-month follow-up visit for safety.
Arm/Group | All Participants
Number analyzed (Participants) | 726
titers
  Serotype 1:Before 13vPnC (Year 5),(n=690) | 10 [8.7 to 10.7]
  Serotype 1: After 13vPnC (Year 5),(n=690) | 173 [153.5 to 195.5]
  Serotype 3: Before 13vPnC (Year 5),(n=699) | 8 [7.6 to 9.2]
  Serotype 3: After 13vPnC (Year 5),(n=699) | 62 [56.6 to 68.0]
  Serotype 4 : Before 13vPnC (Year 5),(n=667) | 88 [73.5 to 106.6]
  Serotype 4 : After 13vPnC (Year 5),(n=667) | 1553 [1426.5 to 1691.4]
  Serotype 5 : Before 13vPnC (Year 5),(n=694) | 16 [13.8 to 18.0]
  Serotype 5 :After 13vPnC (Year 5),(n=694) | 290 [257.8 to 326.4]
  Serotype 6A : Before 13vPnC (Year 5),(n=677) | 173 [144.5 to 206.8]
  Serotype 6A : After 13vPnC (Year 5),(n=677) | 4072 [3684.3 to 4500.2]
  Serotype 6B : Before 13vPnC (Year 5),(n=650) | 209 [174.0 to 252.1]
  Serotype 6B : After 13vPnC (Year 5),(n=650) | 3504 [3181.3 to 3859.7]
  Serotype 7F: Before 13vPnC (Year 5),(n=687) | 122 [100.9 to 147.7]
  Serotype 7F: After 13vPnC (Year 5),(n=687) | 1697 [1569.0 to 1834.7]
  Serotype 9V: Before 13vPnC (Year 5),(n=671) | 97 [78.1 to 119.5]
  Serotype 9V: After 13vPnC (Year 5),(n=671) | 1669 [1479.9 to 1882.6]
  Serotype 14: Before 13vPnC (Year 5),(n=678) | 289 [250.5 to 332.9]
  Serotype 14: After 13vPnC (Year 5),(n=678) | 1096 [1011.1 to 1187.9]
  Serotype 18C: Before 13vPnC (Year 5),(n=683) | 120 [100.5 to 143.6]
  Serotype 18C: After 13vPnC (Year 5),(n=683) | 1748 [1573.5 to 1941.9]
  Serotype 19A: Before 13vPnC (Year 5),(n=696) | 113 [99.0 to 127.9]
  Serotype 19A: After 13vPnC (Year 5),(n=696) | 900 [827.1 to 978.4]
  Serotype 19F: Before 13vPnC (Year 5),(n=649) | 38 [31.5 to 45.1]
  Serotype 19F: After 13vPnC (Year 5),(n=649) | 1146 [1024.6 to 1282.9]
  Serotype 23F: Before 13vPnC (Year 5),(n=685) | 50 [42.2 to 59.0]
  Serotype 23F: After 13vPnC (Year 5),(n=685) | 1819 [1620.2 to 2043.0]

5. Other Pre Specified Outcome: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold-Rises (GMFRs) 1 Month After 13vPnC Re-vaccinated Dose (Year 5) Relative to Before 13vPnC (Year 5)
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined from before 13vPnC (Year 5) to 1 month after 13vPnC re-vaccinated dose (Year 5) and were summarized geometric means and 2-sided 95% CIs, which were computed using the logarithmically transformed assay results. CI for GMFRs were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rises. GMFRs were calculated using all participants with available data from both before 13vPnC (Year 5) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws. n=participants with valid and determinate assay results for the specified serotype from both before 13vPnC (Year 5) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Time Frame: before 13vPnC (Year 5), 1 month after 13vPnC re-vaccinated dose (Year 5)
Population: All-available immunogenicity population at Year 5 included participants who had at least 1 valid and determinate assay result related to the proposed analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rises
Arm/Group | All Participants
Number analyzed (Participants) | 726
fold-rises
  Serotype 1 (n=690) | 18.0 [15.72 to 20.53]
  Serotype 3(n=699) | 7.4 [6.70 to 8.19]
  Serotype 4(n=667) | 17.6 [14.59 to 21.12]
  Serotype 5 (n=694) | 18.4 [16.12 to 20.99]
  Serotype 6A(n=677) | 23.6 [19.74 to 28.11]
  Serotype 6B(n=650) | 16.7 [13.98 to 20.02]
  Serotype 7F(n=687) | 13.9 [11.48 to 16.83]
  Serotype 9V(n=671) | 17.3 [14.10 to 21.17]
  Serotype 14(n=678) | 3.8 [3.32 to 4.34]
  Serotype 18C(n=683) | 14.6 [12.27 to 17.25]
  Serotype 19A(n=696) | 8.0 [7.07 to 9.04]
  Serotype 19F(n=649) | 30.4 [25.47 to 36.34]
  Serotype 23F(n=685) | 36.5 [30.84 to 43.12]

6. Other Pre Specified Outcome: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 1 Month After 13vPnC (Year 0) and 1 Month After 13vPnC Re-vaccinated Dose (Year 5)
Description: Serotype-specific OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of participants using a microcolony OPA (mcOPA) assay. GMTs (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data for 1 month after 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5) blood draws. CI for GMTs were back transformations of a CI based on the Student t distribution for the mean logarithm of the titers. Participants in this population must have immunogenicity data at both the Year 0 and Year 5 time points.n=participants with valid and determinate assay results for the specified serotype for both 1 month after 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Time Frame: 1 month after 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5)
Population: All-available immunogenicity population at Year 0 and 5 included participants who had at least 1 valid and determinate assay result related to the proposed analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | All Participants
Number analyzed (Participants) | 598
titers
  Serotype 1:After 13vPnC (Year 0),(n=381) | 217 [184.0 to 255.0]
  Serotype 1: After 13vPnC (Year 5),(n=381) | 183 [156.6 to 214.6]
  Serotype 3: After 13vPnC (Year 0),(n=374) | 69 [60.0 to 78.7]
  Serotype 3: After 13vPnC (Year 5),(n=374) | 61 [54.4 to 69.0]
  Serotype 4 : After 13vPnC (Year 0),(n=382) | 1905 [1666.7 to 2177.5]
  Serotype 4 : After 13vPnC (Year 5),(n=382) | 1589 [1426.0 to 1771.3]
  Serotype 5 : After 13vPnC (Year 0),(n=374) | 129 [104.5 to 160.1]
  Serotype 5 :After 13vPnC (Year 5),(n=374) | 300 [256.8 to 350.4]
  Serotype 6A : After 13vPnC (Year 0),(n=390) | 2779 [2345.5 to 3293.0]
  Serotype 6A : After 13vPnC (Year 5),(n=390) | 4196 [3677.1 to 4787.1]
  Serotype 6B : After 13vPnC (Year 0),(n=380) | 3089 [2662.6 to 3584.8]
  Serotype 6B : After 13vPnC (Year 5),(n=380) | 3541 [3158.7 to 3968.9]
  Serotype 7F: After 13vPnC (Year 0),(n=372) | 2196 [1839.7 to 2620.3]
  Serotype 7F: After 13vPnC (Year 5),(n=372) | 1768 [1596.9 to 1958.3]
  Serotype 9V: After 13vPnC (Year 0),(n=387) | 1343 [1097.1 to 1643.7]
  Serotype 9V: After 13vPnC (Year 5),(n=387) | 1768 [1501.6 to 2081.6]
  Serotype 14: After 13vPnC (Year 0),(n=383) | 1169 [994.7 to 1374.1]
  Serotype 14: After 13vPnC (Year 5),(n=383) | 1135 [1017.5 to 1265.1]
  Serotype 18C: After 13vPnC (Year 0),(n=381) | 1728 [1420.9 to 2101.1]
  Serotype 18C: After 13vPnC (Year 5),(n=381) | 1772 [1540.0 to 2038.3]
  Serotype 19A: After 13vPnC (Year 0),(n=378) | 879 [769.0 to 1005.4]
  Serotype 19A: After 13vPnC (Year 5),(n=378) | 858 [763.9 to 963.0]
  Serotype 19F: After 13vPnC (Year 0),(n=369) | 472 [383.9 to 579.9]
  Serotype 19F: After 13vPnC (Year 5),(n=369) | 1139 [982.7 to 1319.6]
  Serotype 23F: After 13vPnC (Year 0),(n=368) | 494 [396.4 to 615.2]
  Serotype 23F: After 13vPnC (Year 5),(n=368) | 1955 [1700.6 to 2246.7]

7. Other Pre Specified Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rises (GMFRs) 1 Month After 13vPnC Re-vaccinated Dose (Year 5) Relative to 1 Month After 13vPnC (Year 0)
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined from 1 month after 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5) and were summarized geometric means and 2-sided 95% CIs, which were computed using the logarithmically transformed assay results. CI for GMFRs were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rises. GMFRs were calculated using all participants with available data from both 1 month after 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Time Frame: 1 month after 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5)
Population: All-available immunogenicity population at Years 0 and 5. n=participants with valid and determinate assay results for the specified serotype from both 1 month after 13vPnC (Year 0) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rises
Arm/Group | All Participants
Number analyzed (Participants) | 598
fold-rises
  Serotype 1 (n=381) | 0.8 [0.70 to 1.02]
  Serotype 3(n=374) | 0.9 [0.79 to 1.01]
  Serotype 4(n=382) | 0.8 [0.73 to 0.95]
  Serotype 5 (n=374) | 2.3 [1.92 to 2.80]
  Serotype 6A(n=390) | 1.5 [1.31 to 1.74]
  Serotype 6B(n=380) | 1.1 [1.00 to 1.31]
  Serotype 7F(n=372) | 0.8 [0.67 to 0.96]
  Serotype 9V(n=387) | 1.3 [1.08 to 1.60]
  Serotype 14(n=383) | 1.0 [0.83 to 1.13]
  Serotype 18C(n=381) | 1.0 [0.86 to 1.22]
  Serotype 19A(n=378) | 1.0 [0.88 to 1.08]
  Serotype 19F(n=369) | 2.4 [2.01 to 2.90]
  Serotype 23F(n=368) | 4.0 [3.26 to 4.80]

8. Other Pre Specified Outcome: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) Before 13vPnC (Year 0) and 1 Month After 13vPnC Re-vaccinated Dose (Year 5)
Description: Serotype-specific OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of participants using a microcolony OPA (mcOPA) assay. GMTs (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data for before 13vPnC (Year 0) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws. CI for GMTs were back transformations of a CI based on the Student t distribution for the mean logarithm of the titers. Participants in this population must have immunogenicity data at both the Year 0 and Year 5 time points.
Time Frame: before 13vPnC (Year 0) and 1 month after 13vPnC re-vaccinated dose (Year 5)
Population: All-available immunogenicity population at Years 0 and 5. n=participants with valid and determinate assay results for the specified serotype for both before 13vPnC (Year 0) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | All Participants
Number analyzed (Participants) | 598
titers
  Serotype 1:Before 13vPnC (Year 0),(n=384) | 6 [5.6 to 6.9]
  Serotype 1: After 13vPnC (Year 5),(n=384) | 171 [145.4 to 200.4]
  Serotype 3: Before 13vPnC (Year 0),(n=380) | 6 [5.6 to 6.9]
  Serotype 3: After 13vPnC (Year 5),(n=380) | 60 [53.0 to 67.8]
  Serotype 4 : Before 13vPnC (Year 0),(n=310) | 22 [16.3 to 28.9]
  Serotype 4 : After 13vPnC (Year 5),(n=310) | 1558 [1379.0 to 1761.0]
  Serotype 5 : Before 13vPnC (Year 0),(n=370) | 5 [4.6 to 5.4]
  Serotype 5 :After 13vPnC (Year 5),(n=370) | 284 [241.8 to 333.1]
  Serotype 6A : Before 13vPnC (Year 0),(n=356) | 18 [14.3 to 23.1]
  Serotype 6A : After 13vPnC (Year 5),(n=356) | 4072 [3533.5 to 4692.1]
  Serotype 6B : Before 13vPnC (Year 0),(n=333) | 53 [38.7 to 71.6]
  Serotype 6B : After 13vPnC (Year 5),(n=333) | 3341 [2930.6 to 3809.9]
  Serotype 7F: Before 13vPnC (Year 0),(n=330) | 10 [7.7 to 12.2]
  Serotype 7F: After 13vPnC (Year 5),(n=330) | 1818 [1624.0 to 2035.0]
  Serotype 9V: Before 13vPnC (Year 0),(n=352) | 28 [21.3 to 37.5]
  Serotype 9V: After 13vPnC (Year 5),(n=352) | 1725 [1451.1 to 2050.8]
  Serotype 14: Before 13vPnC (Year 0),(n=369) | 67 [50.8 to 87.2]
  Serotype 14: After 13vPnC (Year 5),(n=369) | 1164 [1041.9 to 1300.8]
  Serotype 18C: Before 13vPnC (Year 0),(n=361) | 20 [15.7 to 25.2]
  Serotype 18C: After 13vPnC (Year 5),(n=361) | 1824 [1579.7 to 2105.6]
  Serotype 19A: Before 13vPnC (Year 0),(n=348) | 28 [22.6 to 33.8]
  Serotype 19A: After 13vPnC (Year 5),(n=348) | 849 [749.6 to 961.0]
  Serotype 19F: Before 13vPnC (Year 0),(n=377) | 14 [11.3 to 16.7]
  Serotype 19F: After 13vPnC (Year 5),(n=377) | 1106 [954.7 to 1281.3]
  Serotype 23F: Before 13vPnC (Year 0),(n=350) | 9 [7.2 to 10.2]
  Serotype 23F: After 13vPnC (Year 5),(n=350) | 1851 [1590.3 to 2155.3]

9. Other Pre Specified Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rises (GMFRs) 1 Month After 13vPnC Re-vaccinated Dose (Year 5) Relative to Before 13vPnC (Year 0)
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined from before13vPnC (Year 0) to 1 month after 13vPnC re-vaccinated dose (Year 5) and were summarized geometric means and 2-sided 95% CIs, which were computed using the logarithmically transformed assay results. CI for GMFRs were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rises. GMFRs were calculated using all participants with available data from both before 13vPnC (Year 0) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Time Frame: before 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5)
Population: All-available immunogenicity population at Years 0 and 5. n=participants with valid and determinate assay results for the specified serotype from both before 13vPnC (Year 0) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rises
Arm/Group | All Participants
Number analyzed (Participants) | 598
fold-rises
  Serotype 1 (n=384) | 27.5 [23.05 to 32.78]
  Serotype 3(n=380) | 9.7 [8.34 to 11.19]
  Serotype 4(n=310) | 71.8 [53.28 to 96.69]
  Serotype 5 (n=370) | 57.0 [48.03 to 67.58]
  Serotype 6A(n=356) | 224.1 [171.09 to 293.51]
  Serotype 6B(n=333) | 63.5 [46.14 to 87.45]
  Serotype 7F(n=330) | 188.0 [147.92 to 238.83]
  Serotype 9V(n=352) | 61.0 [45.19 to 82.31]
  Serotype 14(n=369) | 17.5 [13.40 to 22.86]
  Serotype 18C(n=361) | 91.7 [71.33 to 117.84]
  Serotype 19A(n=348) | 30.7 [24.99 to 37.77]
  Serotype 19F(n=377) | 80.5 [64.90 to 99.92]
  Serotype 23F(n=350) | 216.5 [172.97 to 270.87]

10. Other Pre Specified Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT) Before and 1 Month After 13vPnC (Year 0), 1, 2, 3, 4 Years After Initial Vaccination (Year 0); Before and 1 Month After 13vPnC (Year 5)
Description: Serotype-specific OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of participants using a microcolony OPA (mcOPA) assay. GMT (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data before, 1 month after 13vPnC (Year 0), at Years 1, 2, 3 and 4 after initial vaccination (Year 0), before, 1 month after 13vPnC (Year 5) blood draws. CI for GMT were back transformations of a CI based on the Student t distribution for the mean logarithm of the titers. n=participants with valid and determinate assay results for the specified serotype at before, 1 month after 13vPnC (Year 0), at Years 1, 2, 3 and 4 after initial vaccination (Year 0), before, 1 month after 13vPnC (Year 5) blood draws.
Time Frame: Before,1 month after 13vPnC (Year 0), 1, 2, 3, 4 years after initial vaccination (Year 0); before,1 month after 13vPnC (Year 5)
Population: Subset of all-available immunogenicity population with data at Years 0 through 5 included participants with immunogenicity data at all-time points from Year 0 through Year 5 within the protocol specified time window.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | All Participants
Number analyzed (Participants) | 130
titers
  Serotype 1: Before 13vPnC dose Year 0 (n=92) | 6 [4.9 to 7.0]
  Serotype 1: After 13vPnC dose at Year 0 (n=92) | 200 [143.5 to 278.0]
  Serotype 1: Year 1 (n=125) | 19 [14.0 to 26.7]
  Serotype 1: Year 2 (n=128) | 14 [10.1 to 18.2]
  Serotype 1: Year 3 (n=128) | 11 [8.3 to 14.5]
  Serotype 1: Year 4 (n=127) | 10 [7.4 to 12.4]
  Serotype 1: Before 13vPnC dose Year 5 (n=126) | 10 [7.8 to 12.8]
  Serotype 1: After 13vPnC dose at Year 5 (n=126) | 203 [158.5 to 260.6]
  Serotype 3: Before 13vPnC dose Year 0 (n=90) | 6 [4.9 to 7.3]
  Serotype 3: After 13vPnC dose Year 0 (n=91) | 63 [48.1 to 83.6]
  Serotype 3: Year 1 (n=129) | 14 [10.7 to 17.2]
  Serotype 3: Year 2 (n=129) | 12 [9.2 to 14.7]
  Serotype 3: Year 3 (n=129) | 9 [7.1 to 10.7]
  Serotype 3: Year 4 (n=128) | 9 [7.2 to 11.3]
  Serotype 3: Before 13vPnC dose Year 5 (n=129) | 9 [7.3 to 11.7]
  Serotype 3: After 13vPnC dose at Year 5 (n=128) | 55 [44.6 to 68.1]
  Serotype 4: Before 13vPnC dose Year 0 (n=74) | 16 [8.8 to 27.3]
  Serotype 4: After 13vPnC dose at Year 0 (n=91) | 1896 [1429.7 to 2514.2]
  Serotype 4: Year 1 (n=126) | 442 [309.0 to 632.4]
  Serotype 4: Year 2 (n=121) | 181 [117.1 to 278.7]
  Serotype 4: Year 3 (n=125) | 137 [89.4 to 211.0]
  Serotype 4: Year 4 (n=123) | 97 [62.2 to 151.5]
  Serotype 4: Before 13vPnC dose Year 5 (n=125) | 92 [59.7 to 140.6]
  Serotype 4: After 13vPnC dose at Year 5 (n=128) | 1574 [1340.7 to 1847.9]
  Serotype 5: Before 13vPnC dose Year 0 (n=89) | 5 [4.1 to 5.2]
  Serotype 5: After 13vPnC dose at Year 0 (n=93) | 145 [96.5 to 216.6]
  Serotype 5: Year 1 (n=130) | 32 [22.8 to 43.7]
  Serotype 5: Year 2 (n=128) | 20 [14.4 to 27.0]
  Serotype 5: Year 3 (n=128) | 17 [12.3 to 23.0]
  Serotype 5: Year 4 (n=128) | 14 [10.7 to 19.3]
  Serotype 5: Before 13vPnC dose Year 5 (n=129) | 13 [9.9 to 17.8]
  Serotype 5: After 13vPnC dose at Year 5 (n=128) | 273 [204.7 to 365.2]
  Serotype 6A: Before 13vPnC dose Year 0 (n=87) | 16 [9.9 to 26.1]
  Serotype 6A: After 13vPnC dose Year 0 (n=94) | 2158 [1456.8 to 3196.6]
  Serotype 6A: Year 1 (n=126) | 748 [532.4 to 1051.3]
  Serotype 6A: Year 2 (n=129) | 405 [275.0 to 595.8]
  Serotype 6A: Year 3 (n=127) | 282 [187.7 to 424.1]
  Serotype 6A: Year 4 (n=126) | 203 [134.6 to 306.1]
  Serotype 6A: Before 13vPnC dose Year 5 (n=125) | 166 [107.5 to 255.3]
  Serotype 6A: After 13vPnC dose Year 5 (n=129) | 3777 [2916.3 to 4891.2]
  Serotype 6B: Before 13vPnC dose Year 0 (n=83) | 88 [46.7 to 165.8]
  Serotype 6B: After 13vPnC dose Year 0 (n=93) | 2950 [2110.7 to 4123.5]
  Serotype 6B: Year 1 (n=122) | 765 [562.2 to 1039.9]
  Serotype 6B: Year 2 (n=121) | 505 [353.9 to 720.2]
  Serotype 6B: Year 3 (n=120) | 373 [253.3 to 549.8]
  Serotype 6B: Year 4 (n=115) | 326 [218.2 to 485.9]
  Serotype 6B: Before 13vPnC dose Year 5 (n=123) | 229 [149.1 to 350.3]
  Serotype 6B: After 13vPnC dose Year 5 (n=127) | 3804 [3216.1 to 4499.0]
  Serotype 7F: Before 13vPnC dose Year 0 (n=80) | 13 [7.9 to 23.0]
  Serotype 7F: After 13vPnC dose Year 0 (n=88) | 2265 [1563.6 to 3280.4]
  Serotype 7F: Year 1 (n=129) | 515 [356.6 to 745.1]
  Serotype 7F: Year 2 (n=128) | 279 [182.4 to 426.9]
  Serotype 7F: Year 3 (n=125) | 253 [165.1 to 387.4]
  Serotype 7F: Year 4 (n=127) | 175 [114.3 to 268.6]
  Serotype 7F: Before 13vPnC dose Year 5 (n=124) | 155 [98.7 to 244.5]
  Serotype 7F: After 13vPnC dose Year 5 (n=129) | 1932 [1585.5 to 2353.7]
  Serotype 9V: Before 13vPnC dose Year 0 (n=88) | 17 [9.7 to 28.3]
  Serotype 9V: After 13vPnC dose Year 0 (n=93) | 1202 [795.7 to 1816.4]
  Serotype 9V: Year 1 (n=125) | 276 [173.2 to 440.3]
  Serotype 9V: Year 2 (n=127) | 136 [83.4 to 221.5]
  Serotype 9V: Year 3 (n=128) | 121 [75.2 to 194.7]
  Serotype 9V: Year 4 (n=124) | 66 [39.8 to 108.7]
  Serotype 9V: Before 13vPnC dose Year 5 (n=128) | 86 [53.1 to 139.9]
  Serotype 9V: After 13vPnC dose Year 5 (n=127) | 1572 [1155.4 to 2139.2]
  Serotype 14: Before 13vPnC dose Year 0 (n=87) | 74 [41.7 to 130.1]
  Serotype 14: After 13vPnC dose Year 0 (n=90) | 1436 [1036.7 to 1989.0]
  Serotype 14: Year 1 (n=124) | 541 [394.3 to 741.1]
  Serotype 14: Year 2 (n=125) | 446 [326.5 to 609.0]
  Serotype 14: Year 3 (n=124) | 416 [302.8 to 571.3]
  Serotype 14: Year 4 (n=125) | 341 [241.9 to 481.4]
  Serotype 14: Before 13vPnC dose Year 5 (n=127) | 335 [244.8 to 457.6]
  Serotype 14: After 13vPnC dose Year 5 (n=128) | 1238 [1046.4 to 1464.2]
  Serotype 18C: Before 13vPnC dose Year 0 (n=82) | 18 [11.4 to 29.2]
  Serotype 18C: After 13vPnC dose Year 0 (n=92) | 1189 [766.6 to 1843.2]
  Serotype 18C: Year 1 (n=127) | 301 [206.2 to 440.4]
  Serotype 18C: Year 2 (n=123) | 170 [115.2 to 251.6]
  Serotype 18C: Year 3 (n=129) | 115 [76.7 to 171.2]
  Serotype 18C: Year 4 (n=126) | 102 [67.6 to 154.9]
  Serotype 18C: Before 13vPnC dose Year 5 (n=127) | 99 [65.9 to 148.1]
  Serotype 18C: After 13vPnC dose Year 5 (n=127) | 1580 [1289.0 to 1937.4]
  Serotype 19A: Before 13vPnC dose Year 0 (n=84) | 24 [15.7 to 37.1]
  Serotype 19A: After 13vPnC dose Year 0 (n=92) | 727 [551.4 to 957.4]
  Serotype 19A: Year 1 (n=130) | 193 [145.9 to 255.4]
  Serotype 19A: Year 2 (n=127) | 135 [100.4 to 181.9]
  Serotype 19A: Year 3 (n=129) | 105 [76.6 to 143.3]
  Serotype 19A: Year 4 (n=129) | 97 [72.0 to 131.6]
  Serotype 19A: Before 13vPnC dose Year 5 (n=130) | 97 [71.7 to 132.3]
  Serotype 19A: After 13vPnC dose Year 5 (n=128) | 874 [729.8 to 1046.1]
  Serotype 19F: Before 13vPnC dose Year 0 (n=94) | 14 [9.3 to 21.1]
  Serotype 19F: After 13vPnC dose Year 0 (n=91) | 448 [298.8 to 670.5]
  Serotype 19F: Year 1 (n=124) | 85 [55.7 to 131.0]
  Serotype 19F: Year 2 (n=128) | 44 [28.9 to 67.3]
  Serotype 19F: Year 3 (n=128) | 35 [23.0 to 54.4]
  Serotype 19F: Year 4 (n=125) | 29 [19.2 to 44.0]
  Serotype 19F: Before 13vPnC dose Year 5 (n=125) | 24 [15.9 to 36.1]
  Serotype 19F: After 13vPnC dose Year 5 (n=125) | 1112 [882.3 to 1400.5]
  Serotype 23F: Before 13vPnC dose Year 0 (n=84) | 9 [6.1 to 13.3]
  Serotype 23F: After 13vPnC dose Year 0 (n=89) | 396 [242.7 to 646.6]
  Serotype 23F: Year 1 (n=127) | 116 [78.9 to 171.6]
  Serotype 23F: Year 2 (n=124) | 95 [64.1 to 141.0]
  Serotype 23F: Year 3 (n=128) | 60 [40.4 to 88.0]
  Serotype 23F: Year 4 (n=127) | 54 [36.8 to 78.6]
  Serotype 23F: Before 13vPnC dose Year 5 (n=127) | 48 [33.0 to 71.1]
  Serotype 23F: After 13vPnC dose Year 5 (n=128) | 1642 [1263.2 to 2133.5]

11. Other Pre Specified Outcome: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rises (GMFRs) 1 Month After 13vPnC (Year 0),1, 2, 3, 4 Years After Initial Vaccination (Year 0); Before and 1 Month After 13vPnC (Year 5) Relative to Before 13vPnC (Year 0)
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined from before to 1 month after 13vPnC (Year 0), at years 1, 2, 3 and 4 after initial vaccination (Year 0), before, 1 month after 13vPnC (Year 5) and were summarized geometric means and 2-sided 95% CIs, which were computed using the logarithmically transformed assay results. CI for GMFRs were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rises. GMFRs were calculated using all participants with available data from both the baseline and the various time points.
Time Frame: Before, 1 month after 13vPnC (Year 0), at years 1, 2, 3 and 4 after initial vaccination (Year 0), before, 1 month after 13vPnC (Year 5)
Population: Subset of all-available immunogenicity population with data at Years 0 through 5 included participants with immunogenicity data at all-time points from Year 0 through Year 5 within the protocol specified time window. n=participants with valid and determinate assay results for both the before 13vPnC (Year 0) and all the specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rises
Arm/Group | All Participants
Number analyzed (Participants) | 130
fold-rises
  Serotype 1:After 13vPnC dose at Year 0 (n=89) | 34.0 [24.24 to 47.66]
  Serotype 1: Year 1 (n= 90) | 3.5 [2.45 to 5.00]
  Serotype 1: Year 2 (n=91) | 2.4 [1.72 to 3.26]
  Serotype 1: Year 3 (n= 92) | 1.8 [1.38 to 2.47]
  Serotype 1: Year 4 (n= 90) | 1.6 [1.24 to 2.09]
  Serotype 1: Before 13vPnC dose Year 5 (n=89) | 1.7 [1.26 to 2.16]
  Serotype 1: After 13vPnC dose at Year 5 (n=89) | 39.3 [28.69 to 53.81]
  Serotype 3: After 13vPnC dose at Year 0 (n=87) | 10.4 [7.65 to 14.23]
  Serotype 3: Year 1 (n=89) | 2.0 [1.59 to 2.58]
  Serotype 3: Year 2 (n=89) | 1.6 [1.29 to 2.01]
  Serotype 3: Year 3 (n=89) | 1.3 [1.04 to 1.56]
  Serotype 3: Year 4 (n=89) | 1.4 [1.15 to 1.76]
  Serotype 3: Before 13vPnC dose Year 5 (n=90) | 1.5 [1.14 to 1.86]
  Serotype 3: After 13vPnC dose at Year 5 (n=89) | 9.1 [6.93 to 12.07]
  Serotype 4: After 13vPnC dose at Year 0 (n=72) | 118.9 [65.63 to 215.39]
  Serotype 4: Year 1 (n=74) | 21.3 [11.90 to 38.06]
  Serotype 4: Year 2 (n=71) | 8.3 [4.66 to 14.95]
  Serotype 4: Year 3 (n=70) | 6.5 [3.75 to 11.15]
  Serotype 4: Year 4 (n=71) | 4.6 [2.73 to 7.63]
  Serotype 4: Before 13vPnC dose Year 5 (n=71) | 4.7 [2.80 to 7.74]
  Serotype 4: After 13vPnC dose at Year 5 (n=73) | 98.7 [54.38 to 179.10]
  Serotype 5: After 13vPnC dose at Year 0 (n=87) | 29.5 [19.21 to 45.45]
  Serotype 5: Year 1 (n=89) | 6.1 [4.18 to 8.91]
  Serotype 5: Year 2 (n=88) | 3.7 [2.57 to 5.40]
  Serotype 5: Year 3 (n=88) | 2.9 [2.05 to 4.19]
  Serotype 5: Year 4 (n=88) | 2.6 [1.84 to 3.59]
  Serotype 5: Before 13vPnC dose Year 5 (n=88) | 2.3 [1.67 to 3.29]
  Serotype 5: After 13vPnC dose at Year 5 (n=87) | 60.6 [42.73 to 86.06]
  Serotype 6A: After 13vPnC dose Year 0 (n=86) | 126.8 [69.14 to 232.51]
  Serotype 6A: Year 1 (n=85) | 38.3 [22.35 to 65.79]
  Serotype 6A: Year 2 (n=87) | 21.9 [12.98 to 36.99]
  Serotype 6A: Year 3 (n=86) | 14.8 [8.83 to 24.79]
  Serotype 6A: Year 4 (n=85) | 11.7 [7.00 to 19.62]
  Serotype 6A: Before 13vPnC dose Year 5 (n=85) | 9.2 [5.40 to 15.81]
  Serotype 6A: After 13vPnC dose Year 5 (n=86) | 219.2 [123.97 to 387.54]
  Serotype 6B: After 13vPnC dose Year 0 (n=81) | 33.3 [17.17 to 64.74]
  Serotype 6B: Year 1 (n=78) | 8.9 [4.88 to 16.21]
  Serotype 6B: Year 2 (n=78) | 5.7 [3.18 to 10.14]
  Serotype 6B: Year 3 (n=77) | 4.3 [2.33 to 7.98]
  Serotype 6B: Year 4 (n=73) | 3.3 [1.91 to 5.75]
  Serotype 6B: Before 13vPnC dose Year 5 (n=81) | 2.9 [1.63 to 5.28]
  Serotype 6B: After 13vPnC dose Year 5 (n=81) | 38.8 [19.92 to 75.61]
  Serotype 7F: After 13vPnC dose Year 0 (n=75) | 168.6 [88.78 to 320.29]
  Serotype 7F: Year 1 (n=80) | 37.1 [19.84 to 69.34]
  Serotype 7F: Year 2 (n=78) | 18.7 [10.16 to 34.57]
  Serotype 7F: Year 3 (n=76) | 17.8 [9.69 to 32.66]
  Serotype 7F: Year 4 (n=78) | 10.4 [5.69 to 18.93]
  Serotype 7F: Before 13vPnC dose Year 5 (n=77) | 8.4 [4.57 to 15.56]
  Serotype 7F: After 13vPnC dose Year 5 (n=80) | 163.6 [95.30 to 280.70]
  Serotype 9V: After 13vPnC dose Year 0 (n=86) | 68.2 [37.54 to 123.92]
  Serotype 9V: Year 1 (n=86) | 12.2 [6.94 to 21.55]
  Serotype 9V: Year 2 (n=87) | 5.6 [3.30 to 9.63]
  Serotype 9V: Year 3 (n=88) | 5.3 [3.20 to 8.80]
  Serotype 9V: Year 4 (n=84) | 3.0 [1.79 to 5.00]
  Serotype 9V: Before 13vPnC dose Year 5 (n=87) | 3.8 [2.19 to 6.66]
  Serotype 9V: After 13vPnC dose Year 5 (n=86) | 99.3 [54.99 to 179.41]
  Serotype 14: After 13vPnC dose Year 0 (n=83) | 22.4 [12.42 to 40.22]
  Serotype 14: Year 1 (n=84) | 7.3 [4.35 to 12.22]
  Serotype 14: Year 2 (n=85) | 6.2 [3.86 to 10.11]
  Serotype 14: Year 3 (n=82) | 5.2 [3.12 to 8.80]
  Serotype 14: Year 4 (n=84) | 5.5 [3.26 to 9.42]
  Serotype 14: Before 13vPnC dose Year 5 (n=86) | 4.7 [2.85 to 7.86]
  Serotype 14: After 13vPnC dose Year 5 (n=86) | 19.9 [11.37 to 35.00]
  Serotype 18C: After 13vPnC dose Year 0 (n=79) | 58.2 [31.53 to 107.35]
  Serotype 18C: Year 1 (n=81) | 12.3 [7.45 to 20.29]
  Serotype 18C: Year 2 (n=81) | 6.2 [3.73 to 10.34]
  Serotype 18C: Year 3 (n=81) | 4.5 [2.82 to 7.30]
  Serotype 18C: Year 4 (n=79) | 3.9 [2.46 to 6.22]
  Serotype 18C: Before 13vPnC dose Year 5 (n=81) | 3.9 [2.40 to 6.28]
  Serotype 18C: After 13vPnC dose Year 5 (n=79) | 82.7 [50.04 to 136.70]
  Serotype 19A: After 13vPnC dose Year 0 (n=81) | 28.4 [18.04 to 44.69]
  Serotype 19A: Year 1 (n=84) | 7.3 [4.72 to 11.16]
  Serotype 19A: Year 2 (n=82) | 5.4 [3.55 to 8.18]
  Serotype 19A: Year 3 (n=84) | 4.1 [2.72 to 6.10]
  Serotype 19A: Year 4 (n=84) | 3.7 [2.42 to 5.61]
  Serotype 19A: Before 13vPnC dose Year 5 (n=84) | 3.8 [2.45 to 5.99]
  Serotype 19A: After 13vPnC dose Year 5 (n=83) | 36.4 [23.40 to 56.57]
  Serotype 19F: After 13vPnC dose Year 0 (n=90) | 32.8 [20.67 to 51.98]
  Serotype 19F: Year 1 (n=91) | 6.3 [4.08 to 9.86]
  Serotype 19F: Year 2 (n=93) | 3.9 [2.58 to 6.02]
  Serotype 19F: Year 3 (n=92) | 2.7 [1.76 to 4.09]
  Serotype 19F: Year 4 (n=91) | 2.4 [1.62 to 3.56]
  Serotype 19F: Before 13vPnC dose Year 5 (n=90) | 1.9 [1.26 to 2.83]
  Serotype 19F: After 13vPnC dose Year 5 (n=89) | 81.6 [52.36 to 127.08]
  Serotype 23F: After 13vPnC dose Year 0 (n=79) | 41.2 [23.36 to 72.69]
  Serotype 23F: Year 1 (n=84) | 12.6 [7.69 to 20.62]
  Serotype 23F: Year 2 (n=81) | 9.6 [5.81 to 15.78]
  Serotype 23F: Year 3 (n=84) | 6.6 [4.13 to 10.41]
  Serotype 23F: Year 4 (n=84) | 5.8 [3.68 to 9.26]
  Serotype 23F: Before 13vPnC dose Year 5 (n=83) | 5.3 [3.31 to 8.53]
  Serotype 23F: After 13vPnC dose Year 5 (n=82) | 194.0 [115.99 to 324.32]

12. Other Pre Specified Outcome: Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentration (GMCs) 1 Month After 13vPnC (Year 5)
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) for adult participants are presented. GMC (13vPnC) and corresponding 2-sided 95 percent (%) CIs were evaluated. Geometric means were calculated using all participants with available data for 1 month after 13vPnC Dose 1 blood draw. CI for GMC are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: 1 month after 13vPnC (Year 5)
Population: All-available immunogenicity population at Year 5. n=participants with valid and determinate assay results for the specified serotype at 1 month after 13vPnC (Year 5) blood draws for each treatment arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter(mcg/mL)
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 363 | 363
microgram per milliliter(mcg/mL)
  Serotype 1 (n=357, 345) | 5.92 [5.33 to 6.57] | 5.83 [5.20 to 6.55]
  Serotype 3(n=343, 338) | 0.69 [0.62 to 0.76] | 0.72 [0.65 to 0.80]
  Serotype 4(n=357,345) | 4.90 [4.42 to 5.44] | 4.77 [4.22 to 5.39]
  Serotype 5(n=357,345) | 7.49 [6.71 to 8.35] | 8.02 [7.16 to 8.99]
  Serotype 6A(n=357,345) | 13.59 [12.01 to 15.39] | 13.45 [11.67 to 15.51]
  Serotype 6B(n=355,345) | 20.18 [17.74 to 22.96] | 21.76 [18.97 to 24.96]
  Serotype 7F(n=357,345) | 8.48 [7.72 to 9.30] | 8.70 [7.91 to 9.58]
  Serotype 9V(n=357,345) | 5.91 [5.37 to 6.51] | 6.35 [5.74 to 7.02]
  Serotype 14(n=357,345) | 15.57 [13.94 to 17.39] | 16.39 [14.70 to 18.28]
  Serotype 18C(n=357,345) | 7.77 [7.06 to 8.55] | 8.46 [7.58 to 9.44]
  Serotype 19A(n=357,345) | 16.77 [15.09 to 18.64] | 17.97 [16.14 to 20.01]
  Serotype 19F(n=357,345) | 16.83 [14.86 to 19.06] | 18.18 [15.77 to 20.96]
  Serotype 23F(n=357,345) | 18.15 [15.87 to 20.76] | 20.25 [17.57 to 23.32]
Statistical Analysis 1: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Geometric Mean Ratio = 1.01, 95% CI 2-sided [0.87 to 1.18]
Statistical Analysis 2: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; Geometric Mean Ratio = 0.95, 95% CI 2-sided [0.82 to 1.10]
Statistical Analysis 3: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; Geometric Mean Ratio = 1.03, 95% CI 2-sided [0.88 to 1.21]
Statistical Analysis 4: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; Geometric Mean Ratio = 0.93, 95% CI 2-sided [0.80 to 1.09]
Statistical Analysis 5: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; Geometric Mean Ratio = 1.01, 95% CI 2-sided [0.84 to 1.22]
Statistical Analysis 6: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; Geometric Mean Ratio = 0.93, 95% CI 2-sided [0.77 to 1.12]
Statistical Analysis 7: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; Geometric Mean Ratio = 0.97, 95% CI 2-sided [0.85 to 1.11]
Statistical Analysis 8: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; Geometric Mean Ratio = 0.93, 95% CI 2-sided [0.81 to 1.07]
Statistical Analysis 9: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; Geometric Mean Ratio = 0.95, 95% CI 2-sided [0.81 to 1.11]
Statistical Analysis 10: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; Geometric Mean Ratio = 0.92, 95% CI 2-sided [0.79 to 1.06]
Statistical Analysis 11: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; Geometric Mean Ratio = 0.93, 95% CI 2-sided [0.80 to 1.08]
Statistical Analysis 12: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 12]; Test type: Superiority or Other; Geometric Mean Ratio = 0.93, 95% CI 2-sided [0.77 to 1.12]
Statistical Analysis 13: Comparison: 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) vs Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5); [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; Geometric Mean Ratio = 0.90, 95% CI 2-sided [0.74 to 1.09]

13. Other Pre Specified Outcome: Serotype-specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentration (GMCs) Before 13vPnC (Year 5) and 1 Month After 13vPnC Re-vaccinated Dose (Year 5)
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) for adult participants are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data before 13vPnC (Year 5) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draw. CI for GMC are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations. Participants in this population must have immunogenicity data at both Year 5 time points.
Time Frame: before 13vPnC (Year 5) and 1 month after 13vPnC re-vaccinated dose (Year 5)
Population: All-available immunogenicity population at Year 5. n=participants with valid and determinate assay results for the specified serotype at before 13vPnC (Year 5) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | All Participants
Number analyzed (Participants) | 726
mcg/mL
  Serotype 1:Before 13vPnC (Year 5),(n=665) | 1.27 [1.16 to 1.40]
  Serotype 1: After 13vPnC (Year 5),(n=665) | 5.87 [5.42 to 6.36]
  Serotype 3: Before 13vPnC (Year 5),(n=623) | 0.33 [0.30 to 0.37]
  Serotype 3: After 13vPnC (Year 5),(n=623) | 0.71 [0.65 to 0.76]
  Serotype 4 : Before 13vPnC (Year 5),(n=663) | 0.67 [0.60 to 0.74]
  Serotype 4 : After 13vPnC (Year 5),(n=663) | 4.83 [4.45 to 5.24]
  Serotype 5 : Before 13vPnC (Year 5),(n=671) | 2.65 [2.45 to 2.87]
  Serotype 5 :After 13vPnC (Year 5),(n=671) | 7.76 [7.16 to 8.41]
  Serotype 6A : Before 13vPnC (Year 5),(n=671) | 2.52 [2.33 to 2.73]
  Serotype 6A : After 13vPnC (Year 5),(n=671) | 13.51 [12.28 to 14.86]
  Serotype 6B : Before 13vPnC (Year 5),(n=668) | 3.12 [2.86 to 3.41]
  Serotype 6B : After 13vPnC (Year 5),(n=668) | 21.04 [19.12 to 23.16]
  Serotype 7F: Before 13vPnC (Year 5),(n=671) | 2.52 [2.31 to 2.76]
  Serotype 7F: After 13vPnC (Year 5),(n=671) | 8.72 [8.16 to 9.33]
  Serotype 9V: Before 13vPnC (Year 5),(n=672) | 2.11 [1.96 to 2.28]
  Serotype 9V: After 13vPnC (Year 5),(n=672) | 6.14 [5.71 to 6.59]
  Serotype 14: Before 13vPnC (Year 5),(n=672) | 5.17 [4.69 to 5.70]
  Serotype 14: After 13vPnC (Year 5),(n=672) | 16.26 [15.03 to 17.58]
  Serotype 18C: Before 13vPnC (Year 5),(n=672) | 2.55 [2.34 to 2.78]
  Serotype 18C: After 13vPnC (Year 5),(n=672) | 8.10 [7.52 to 8.72]
  Serotype 19A: Before 13vPnC (Year 5),(n=671) | 5.47 [5.07 to 5.89]
  Serotype 19A: After 13vPnC (Year 5),(n=671) | 17.29 [16.03 to 18.65]
  Serotype 19F: Before 13vPnC (Year 5),(n=664) | 2.24 [2.02 to 2.47]
  Serotype 19F: After 13vPnC (Year 5),(n=664) | 17.73 [16.10 to 19.53]
  Serotype 23F: Before 13vPnC (Year 5),(n=671) | 2.50 [2.29 to 2.73]
  Serotype 23F: After 13vPnC (Year 5),(n=671) | 19.23 [17.45 to 21.20]

14. Other Pre Specified Outcome: Serotype-specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Fold Rises (GMFRs) 1 Month After 13vPnC Re-vaccinated Dose (Year 5) Relative to Before 13vPnC (Year 5)
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined from before 13vPnC (Year 5) to 1 month after 13vPnC re-vaccinated dose (Year 5) and were summarized geometric means and 2-sided 95% CIs, which were computed using the logarithmically transformed assay results. CI for GMFRs were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rises. GMFRs were calculated using all participants with available data from both before 13vPnC (Year 5) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Time Frame: before 13vPnC (Year 5), 1 month after 13vPnC re-vaccinated dose (Year 5)
Population: All-available immunogenicity population at Year 5. n=participants with valid and determinate assay results for the specified serotype for both before 13vPnC (Year 5) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rises
Arm/Group | All Participants
Number analyzed (Participants) | 726
fold-rises
  Serotype 1 (n=665) | 4.62 [4.22 to 5.05]
  Serotype 3(n=623) | 2.11 [1.99 to 2.24]
  Serotype 4(n=663) | 7.24 [6.60 to 7.95]
  Serotype 5 (n=671) | 2.93 [2.75 to 3.12]
  Serotype 6A(n=671) | 5.35 [4.92 to 5.82]
  Serotype 6B(n=668) | 6.74 [6.19 to 7.34]
  Serotype 7F(n=671) | 3.46 [3.20 to 3.74]
  Serotype 9V(n=672) | 2.90 [2.74 to 3.08]
  Serotype 14(n=672) | 3.14 [2.89 to 3.42]
  Serotype 18C(n=672) | 3.18 [2.96 to 3.41]
  Serotype 19A(n=671) | 3.16 [2.95 to 3.39]
  Serotype 19F(n=664) | 7.93 [7.21 to 8.72]
  Serotype 23F(n=671) | 7.69 [7.05 to 8.39]

15. Other Pre Specified Outcome: Serotype-specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentration (GMCs) 1 Month After 13vPnC (Year 0) and 1 Month After 13vPnC Re-vaccinated Dose (Year 5)
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) for adult participants are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data 1 month after 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5) blood draw. CI for GMC are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations. Participants in this population must have immunogenicity data at both the Year 0 and Year 5 time points
Time Frame: 1 month after 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5)
Population: All-available immunogenicity population at Years 0 and 5. n=participants with valid and determinate assay results for the specified serotype for both 1 month after 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | All Participants
Number analyzed (Participants) | 598
mcg/mL
  Serotype 1:After 13vPnC (Year 0),(n=389) | 4.77 [4.10 to 5.54]
  Serotype 1: After 13vPnC (Year 5),(n=389) | 5.88 [5.32 to 6.50]
  Serotype 3: After 13vPnC (Year 0),(n=378) | 1.26 [1.13 to 1.40]
  Serotype 3: After 13vPnC (Year 5),(n=378) | 0.74 [0.67 to 0.81]
  Serotype 4 : After 13vPnC (Year 0),(n=387) | 2.90 [2.51 to 3.36]
  Serotype 4 : After 13vPnC (Year 5),(n=387) | 5.13 [4.64 to 5.68]
  Serotype 5 : After 13vPnC (Year 0),(n=390) | 6.52 [5.72 to 7.44]
  Serotype 5 :After 13vPnC (Year 5),(n=390) | 8.25 [7.40 to 9.20]
  Serotype 6A : After 13vPnC (Year 0),(n=390) | 6.13 [5.41 to 6.94]
  Serotype 6A : After 13vPnC (Year 5),(n=390) | 13.52 [11.94 to 15.31]
  Serotype 6B : After 13vPnC (Year 0),(n=390) | 8.87 [7.77 to 10.14]
  Serotype 6B : After 13vPnC (Year 5),(n=390) | 20.70 [18.31 to 23.39]
  Serotype 7F: After 13vPnC (Year 0),(n=390) | 9.24 [8.16 to 10.47]
  Serotype 7F: After 13vPnC (Year 5),(n=390) | 8.40 [7.68 to 9.19]
  Serotype 9V: After 13vPnC (Year 0),(n=391) | 5.83 [5.17 to 6.56]
  Serotype 9V: After 13vPnC (Year 5),(n=391) | 6.07 [5.53 to 6.65]
  Serotype 14: After 13vPnC (Year 0),(n=391) | 11.98 [10.33 to 13.91]
  Serotype 14: After 13vPnC (Year 5),(n=391) | 15.04 [13.57 to 16.66]
  Serotype 18C: After 13vPnC (Year 0),(n=390) | 11.64 [10.20 to 13.29]
  Serotype 18C: After 13vPnC (Year 5),(n=390) | 8.25 [7.47 to 9.12]
  Serotype 19A: After 13vPnC (Year 0),(n=391) | 17.43 [15.51 to 19.59]
  Serotype 19A: After 13vPnC (Year 5),(n=391) | 18.48 [16.68 to 20.48]
  Serotype 19F: After 13vPnC (Year 0),(n=388) | 6.56 [5.66 to 7.60]
  Serotype 19F: After 13vPnC (Year 5),(n=388) | 18.26 [16.14 to 20.66]
  Serotype 23F: After 13vPnC (Year 0),(n=391) | 8.03 [6.91 to 9.32]
  Serotype 23F: After 13vPnC (Year 5),(n=391) | 20.17 [17.81 to 22.83]

16. Other Pre Specified Outcome: Serotype-specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Fold Rises (GMFRs) 1 Month After 13vPnC Re-vaccinated Dose (Year 5) Relative to 1 Month After 13vPnC (Year 0)
Description: as for outcome 7
Time Frame: 1 month after 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rises
Arm/Group | All Participants
Number analyzed (Participants) | 598
fold-rises
  Serotype 1 (n=389) | 1.23 [1.07 to 1.42]
  Serotype 3(n=378) | 0.59 [0.54 to 0.64]
  Serotype 4(n=387) | 1.77 [1.56 to 2.01]
  Serotype 5 (n=390) | 1.26 [1.14 to 1.41]
  Serotype 6A(n=390) | 2.21 [1.97 to 2.47]
  Serotype 6B(n=390) | 2.33 [2.08 to 2.61]
  Serotype 7F(n=390) | 0.91 [0.81 to 1.02]
  Serotype 9V(n=391) | 1.04 [0.95 to 1.14]
  Serotype 14(n=391) | 1.25 [1.10 to 1.43]
  Serotype 18C(n=390) | 0.71 [0.64 to 0.79]
  Serotype 19A(n=391) | 1.06 [0.96 to 1.17]
  Serotype 19F(n=388) | 2.78 [2.44 to 3.17]
  Serotype 23F(n=391) | 2.51 [2.23 to 2.83]

17. Other Pre Specified Outcome: Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentration (GMCs) Before 13vPnC (Year 0) and 1 Month After 13vPnC Re-vaccinated Dose (Year 5)
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) for adult participants are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data before 13vPnC (Year 0) and 1 month after 13vPnC re-vaccinated dose (Year 5) blood draw. CI for GMC are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations. Participants in this population must have immunogenicity data at both the Year 0 and Year 5 time points.
Time Frame: before 13vPnC (Year 0) and 1 month after 13vPnC re-vaccinated dose (Year 5)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | All Participants
Number analyzed (Participants) | 598
mcg/mL
  Serotype 1:Before 13vPnC (Year 0),(n=380) | 0.44 [0.38 to 0.50]
  Serotype 1: After 13vPnC (Year 5),(n=380) | 5.86 [5.29 to 6.48]
  Serotype 3: Before 13vPnC (Year 0),(n=368) | 0.47 [0.42 to 0.53]
  Serotype 3: After 13vPnC (Year 5),(n=368) | 0.74 [0.67 to 0.81]
  Serotype 4 : Before 13vPnC (Year 0),(n=373) | 0.22 [0.19 to 0.26]
  Serotype 4 : After 13vPnC (Year 5),(n=373) | 5.21 [4.71 to 5.77]
  Serotype 5 : Before 13vPnC (Year 0),(n=387) | 1.79 [1.65 to 1.95]
  Serotype 5 :After 13vPnC (Year 5),(n=387) | 8.32 [7.46 to 9.27]
  Serotype 6A : Before 13vPnC (Year 0),(n=386) | 1.56 [1.42 to 1.71]
  Serotype 6A : After 13vPnC (Year 5),(n=386) | 13.63 [12.03 to 15.45]
  Serotype 6B : Before 13vPnC (Year 0),(n=383) | 1.76 [1.58 to 1.96]
  Serotype 6B : After 13vPnC (Year 5),(n=383) | 21.09 [18.66 to 23.84]
  Serotype 7F: Before 13vPnC (Year 0),(n=384) | 0.70 [0.62 to 0.79]
  Serotype 7F: After 13vPnC (Year 5),(n=384) | 8.41 [7.70 to 9.19]
  Serotype 9V: Before 13vPnC (Year 0),(n=387) | 0.87 [0.79 to 0.96]
  Serotype 9V: After 13vPnC (Year 5),(n=387) | 6.07 [5.53 to 6.66]
  Serotype 14: Before 13vPnC (Year 0),(n=389) | 1.95 [1.69 to 2.26]
  Serotype 14: After 13vPnC (Year 5),(n=389) | 14.98 [13.51 to 16.61]
  Serotype 18C: Before 13vPnC (Year 0),(n=388) | 0.82 [0.72 to 0.94]
  Serotype 18C: After 13vPnC (Year 5),(n=388) | 8.24 [7.45 to 9.11]
  Serotype 19A: Before 13vPnC (Year 0),(n=388) | 2.92 [2.66 to 3.22]
  Serotype 19A: After 13vPnC (Year 5),(n=388) | 18.52 [16.71 to 20.53]
  Serotype 19F: Before 13vPnC (Year 0),(n=371) | 1.17 [1.03 to 1.33]
  Serotype 19F: After 13vPnC (Year 5),(n=371) | 18.68 [16.46 to 21.19]
  Serotype 23F: Before 13vPnC (Year 0),(n=382) | 0.97 [0.86 to 1.09]
  Serotype 23F: After 13vPnC (Year 5),(n=382) | 20.53 [18.14 to 23.23]

18. Other Pre Specified Outcome: Serotype-specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Fold Rises (GMFRs) 1 Month After 13vPnC Re-vaccinated Dose (Year 5) Relative to Before 13vPnC (Year 0)
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined from Before 13vPnC (Year 0) to 1 month after 13vPnC re-vaccinated dose (Year 5) and were summarized geometric means and 2-sided 95% CIs, which were computed using the logarithmically transformed assay results. CI for GMFRs were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rises. GMFRs were calculated using all participants with available data from both before 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Time Frame: Before 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5)
Population: All-available immunogenicity population at Years 0 and 5. n=participants with valid and determinate assay results for the specified serotype for both before 13vPnC (Year 0),1 month after 13vPnC re-vaccinated dose (Year 5) blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rises
Arm/Group | All Participants
Number analyzed (Participants) | 598
fold-rises
  Serotype 1 (n=380) | 13.37 [11.66 to 15.33]
  Serotype 3(n=368) | 1.57 [1.43 to 1.73]
  Serotype 4(n=373) | 23.59 [20.21 to 27.55]
  Serotype 5 (n=387) | 4.64 [4.17 to 5.16]
  Serotype 6A(n=386) | 8.74 [7.63 to 10.00]
  Serotype 6B(n=383) | 11.96 [10.46 to 13.68]
  Serotype 7F(n=384) | 11.96 [10.53 to 13.57]
  Serotype 9V(n=387) | 6.97 [6.29 to 7.73]
  Serotype 14(n=389) | 7.68 [6.62 to 8.92]
  Serotype 18C(n=388) | 10.04 [8.84 to 11.40]
  Serotype 19A(n=388) | 6.33 [5.66 to 7.09]
  Serotype 19F(n=371) | 15.95 [13.69 to 18.57]
  Serotype 23F(n=382) | 21.18 [18.50 to 24.25]

19. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Before and 1 Month After 13vPnC (Year 0), 1, 2, 3, 4 Years After Initial Vaccination (Year 0); Before and 1 Month After 13vPnC (Year 5)
Description: Participants received either 0.5 mL dose of 13vPnC intramuscular injection into the deltoid muscle of the left arm along with 0.5-mL TIV intramuscular injection into the deltoid muscle of the right arm at Year 0 on Day 1(Dose1, 13vPnC+TIV), or placebo matched to 13vPnC intramuscular injection into the deltoid muscle of the left arm along with 0.5-mL TIV intramuscular injection into the deltoid muscle of the right arm at Year 0 on Day 1(Dose 1, placebo+TIV). Placebo matched to 13vPnC was administered 1 month after(Dose 2, placebo), or 13vPnC was administered 1 month after (Dose 2, 13vPnC).Participants were further followed-up for 1 month,then attended a 6-month follow-up visit for safety.Participants were then followed-up yearly for 4 years.Participants then received 0.5 mL dose of 13vPnC intramuscular injection into the deltoid muscle of the left arm 5 years after initial vaccination.Participants were further followed-up for 1 month, then attended a 6-month follow-up visit for safety.
Time Frame: as for outcome 10
Population: Subset of all-available immunogenicity population with data at Years 0 through 5 included participants with immunogenicity data at all-time points from Years 0 through Year 5 within the protocol specified time window. Here, n=number of participants with valid and determinate assay results for the specified serotype at the given time points.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | All Participants
Number analyzed (Participants) | 130
mcg/mL
  Serotype 1: Before 13vPnC dose Year 0 (n=79) | 0.37 [0.28 to 0.49]
  Serotype 1: After 13vPnC dose at Year 0 (n=83) | 4.53 [3.33 to 6.18]
  Serotype 1: Year 1 (n=119) | 1.96 [1.55 to 2.48]
  Serotype 1: Year 2 (n=124) | 1.56 [1.25 to 1.96]
  Serotype 1: Year 3 (n=126) | 1.34 [1.08 to 1.66]
  Serotype 1: Year 4 (n=125) | 1.32 [1.06 to 1.63]
  Serotype 1: Before 13vPnC dose Year 5 (n=125) | 1.18 [0.95 to 1.47]
  Serotype 1: After 13vPnC dose at Year 5 (n=125) | 6.08 [5.20 to 7.11]
  Serotype 3: Before 13vPnC dose Year 0 (n=81) | 0.42 [0.33 to 0.53]
  Serotype 3: After 13vPnC dose Year 0 (n=82) | 1.15 [0.92 to 1.44]
  Serotype 3: Year 1 (n=115) | 0.37 [0.30 to 0.46]
  Serotype 3: Year 2 (n=122) | 0.34 [0.27 to 0.42]
  Serotype 3: Year 3 (n=119) | 0.30 [0.25 to 0.37]
  Serotype 3: Year 4 (n=117) | 0.31 [0.25 to 0.38]
  Serotype 3: Before 13vPnC dose Year 5 (n=117) | 0.30 [0.24 to 0.38]
  Serotype 3: After 13vPnC dose at Year 5 (n=121) | 0.66 [0.55 to 0.79]
  Serotype 4: Before 13vPnC dose Year 0 (n=80) | 0.19 [0.14 to 0.25]
  Serotype 4: After 13vPnC dose at Year 0 (n=82) | 2.41 [1.74 to 3.35]
  Serotype 4: Year 1 (n=118) | 0.98 [0.77 to 1.26]
  Serotype 4: Year 2 (n=123) | 0.77 [0.61 to 0.98]
  Serotype 4: Year 3 (n=125) | 0.67 [0.53 to 0.85]
  Serotype 4: Year 4 (n=125) | 0.64 [0.50 to 0.82]
  Serotype 4: Before 13vPnC dose Year 5 (n=122) | 0.58 [0.46 to 0.74]
  Serotype 4: After 13vPnC dose at Year 5 (n=125) | 4.62 [3.92 to 5.45]
  Serotype 5: Before 13vPnC dose Year 0 (n=82) | 1.40 [1.17 to 1.69]
  Serotype 5: After 13vPnC dose at Year 0 (n=83) | 5.80 [4.40 to 7.64]
  Serotype 5: Year 1 (n=118) | 3.10 [2.58 to 3.73]
  Serotype 5: Year 2 (n=124) | 2.62 [2.19 to 3.14]
  Serotype 5: Year 3 (n=126) | 2.40 [2.01 to 2.86]
  Serotype 5: Year 4 (n=125) | 2.44 [2.05 to 2.91]
  Serotype 5: Before 13vPnC dose Year 5 (n=125) | 2.41 [2.01 to 2.88]
  Serotype 5: After 13vPnC dose at Year 5 (n=125) | 7.14 [5.95 to 8.57]
  Serotype 6A: Before 13vPnC dose Year 0 (n=82) | 1.34 [1.09 to 1.66]
  Serotype 6A: After 13vPnC dose Year 0 (n=83) | 5.74 [4.29 to 7.68]
  Serotype 6A: Year 1 (n=119) | 3.64 [2.95 to 4.50]
  Serotype 6A: Year 2 (n=124) | 3.10 [2.54 to 3.79]
  Serotype 6A: Year 3 (n=126) | 2.76 [2.26 to 3.38]
  Serotype 6A: Year 4 (n=126) | 2.74 [2.26 to 3.32]
  Serotype 6A: Before 13vPnC dose Year 5 (n=125) | 2.63 [2.16 to 3.21]
  Serotype 6A: After 13vPnC dose Year 5 (n=125) | 14.31 [11.43 to 17.93]
  Serotype 6B: Before 13vPnC dose Year 0 (n=81) | 1.56 [1.23 to 1.97]
  Serotype 6B: After 13vPnC dose Year 0 (n=83) | 8.24 [6.17 to 11.00]
  Serotype 6B: Year 1 (n=119) | 4.96 [3.97 to 6.20]
  Serotype 6B: Year 2 (n=124) | 3.97 [3.23 to 4.88]
  Serotype 6B: Year 3 (n=126) | 3.58 [2.91 to 4.41]
  Serotype 6B: Year 4 (n=126) | 3.53 [2.88 to 4.31]
  Serotype 6B: Before 13vPnC dose Year 5 (n=125) | 3.18 [2.56 to 3.93]
  Serotype 6B: After 13vPnC dose Year 5 (n=124) | 21.61 [17.55 to 26.60]
  Serotype 7F: Before 13vPnC dose Year 0 (n=81) | 0.64 [0.51 to 0.81]
  Serotype 7F: After 13vPnC dose Year 0 (n=83) | 9.14 [6.78 to 12.31]
  Serotype 7F: Year 1 (n=119) | 3.82 [3.05 to 4.79]
  Serotype 7F: Year 2 (n=124) | 3.10 [2.46 to 3.89]
  Serotype 7F: Year 3 (n=126) | 2.58 [2.08 to 3.19]
  Serotype 7F: Year 4 (n=126) | 2.55 [2.05 to 3.18]
  Serotype 7F: Before 13vPnC dose Year 5 (n=124) | 2.36 [1.90 to 2.93]
  Serotype 7F: After 13vPnC dose Year 5 (n=125) | 8.05 [6.68 to 9.71]
  Serotype 9V: Before 13vPnC dose Year 0 (n=80) | 0.77 [0.63 to 0.95]
  Serotype 9V: After 13vPnC dose Year 0 (n=83) | 4.58 [3.62 to 5.81]
  Serotype 9V: Year 1 (n=119) | 2.84 [2.39 to 3.37]
  Serotype 9V: Year 2 (n=124) | 2.37 [1.99 to 2.81]
  Serotype 9V: Year 3 (n=126) | 2.16 [1.82 to 2.56]
  Serotype 9V: Year 4 (n=126) | 2.09 [1.76 to 2.47]
  Serotype 9V: Before 13vPnC dose Year 5 (n=125) | 1.97 [1.67 to 2.34]
  Serotype 9V: After 13vPnC dose Year 5 (n=125) | 5.99 [5.14 to 6.98]
  Serotype 14: Before 13vPnC dose Year 0 (n=82) | 2.21 [1.64 to 2.97]
  Serotype 14: After 13vPnC dose Year 0 (n=83) | 14.48 [10.72 to 19.57]
  Serotype 14: Year 1 (n=119) | 7.71 [6.07 to 9.80]
  Serotype 14: Year 2 (n=124) | 6.82 [5.47 to 8.49]
  Serotype 14: Year 3 (n=126) | 5.71 [4.50 to 7.25]
  Serotype 14: Year 4 (n=126) | 5.31 [4.22 to 6.69]
  Serotype 14: Before 13vPnC dose Year 5 (n=125) | 5.30 [4.20 to 6.70]
  Serotype 14: After 13vPnC dose Year 5 (n=125) | 16.85 [14.07 to 20.18]
  Serotype 18C: Before 13vPnC dose Year 0 (n=82) | 0.81 [0.62 to 1.07]
  Serotype 18C: After 13vPnC dose Year 0 (n=83) | 8.11 [6.03 to 10.89]
  Serotype 18C: Year 1 (n=119) | 3.45 [2.85 to 4.18]
  Serotype 18C: Year 2 (n=124) | 2.82 [2.35 to 3.38]
  Serotype 18C: Year 3 (n=126) | 2.38 [1.98 to 2.86]
  Serotype 18C: Year 4 (n=126) | 2.44 [2.07 to 2.88]
  Serotype 18C: Before 13vPnC dose Year 5 (n=125) | 2.26 [1.89 to 2.71]
  Serotype 18C: After 13vPnC dose Year 5 (n=125) | 6.94 [5.92 to 8.12]
  Serotype 19A: Before 13vPnC dose Year 0 (n=82) | 2.57 [2.13 to 3.11]
  Serotype 19A: After 13vPnC dose Year 0 (n=83) | 14.11 [11.28 to 17.64]
  Serotype 19A: Year 1 (n=119) | 6.95 [5.78 to 8.35]
  Serotype 19A: Year 2 (n=124) | 6.13 [5.19 to 7.25]
  Serotype 19A: Year 3 (n=126) | 5.60 [4.73 to 6.63]
  Serotype 19A: Year 4 (n=126) | 5.47 [4.65 to 6.45]
  Serotype 19A: Before 13vPnC dose Year 5 (n=125) | 5.11 [4.32 to 6.05]
  Serotype 19A: After 13vPnC dose Year 5 (n=125) | 15.77 [13.25 to 18.78]
  Serotype 19F: Before 13vPnC dose Year 0 (n=78) | 0.99 [0.75 to 1.29]
  Serotype 19F: After 13vPnC dose Year 0 (n=83) | 5.64 [4.16 to 7.66]
  Serotype 19F: Year 1 (n=118) | 2.87 [2.29 to 3.60]
  Serotype 19F: Year 2 (n=121) | 2.55 [2.05 to 3.16]
  Serotype 19F: Year 3 (n=124) | 2.28 [1.84 to 2.83]
  Serotype 19F: Year 4 (n=125) | 2.26 [1.83 to 2.81]
  Serotype 19F: Before 13vPnC dose Year 5 (n=123) | 2.10 [1.66 to 2.66]
  Serotype 19F: After 13vPnC dose Year 5 (n=125) | 17.37 [14.23 to 21.20]
  Serotype 23F: Before 13vPnC dose Year 0 (n=80) | 0.97 [0.73 to 1.30]
  Serotype 23F: After 13vPnC dose Year 0 (n=83) | 6.06 [4.38 to 8.39]
  Serotype 23F: Year 1 (n=118) | 3.65 [2.96 to 4.51]
  Serotype 23F: Year 2 (n=123) | 2.93 [2.40 to 3.57]
  Serotype 23F: Year 3 (n=126) | 2.67 [2.19 to 3.25]
  Serotype 23F: Year 4 (n=126) | 2.62 [2.16 to 3.17]
  Serotype 23F: Before 13vPnC dose Year 5 (n=125) | 2.50 [2.05 to 3.04]
  Serotype 23F: After 13vPnC dose Year 5 (n=125) | 16.95 [13.73 to 20.91]

20. Other Pre Specified Outcome: Serotype-specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Fold Rises (GMFRs) 1 Month After 13vPnC (Year 0),1, 2, 3, 4 Years After Initial Vaccination (Year 0); Before and 1 Month After 13vPnC (Year 5) Relative to Before 13vPnC (Year 0)
Description: as for outcome 11
Time Frame: as for outcome 11
Population: Subset of all-available immunogenicity population with data at Years 0 through 5 included participants with immunogenicity data at all-time points from Year 0 through Year 5 within the protocol specified time window. n=participants with valid and determinate assay results for both the before 13vPnC (Year 0) and the specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rises
Arm/Group | All Participants
Number analyzed (Participants) | 130
fold-rises
  Serotype 1:After 13vPnC dose at Year 0 (n=79) | 12.50 [9.25 to 16.90]
  Serotype 1: Year 1 (n=72) | 5.64 [4.32 to 7.35]
  Serotype 1: Year 2 (n=75) | 4.73 [3.73 to 6.00]
  Serotype 1: Year 3 (n=76) | 4.01 [3.15 to 5.11]
  Serotype 1: Year 4 (n=75) | 3.79 [3.00 to 4.78]
  Serotype 1: Before 13vPnC dose Year 5 (n=76) | 3.41 [2.72 to 4.28]
  Serotype 1: After 13vPnC dose at Year 5 (n=77) | 15.25 [11.63 to 19.99]
  Serotype 3: After 13vPnC dose at Year 0 (n=80) | 2.69 [2.21 to 3.28]
  Serotype 3: Year 1 (n=73) | 0.89 [0.74 to 1.07]
  Serotype 3: Year 2 (n=77) | 0.77 [0.66 to 0.90]
  Serotype 3: Year 3 (n= 77) | 0.72 [0.62 to 0.84]
  Serotype 3: Year 4 (n=72) | 0.69 [0.58 to 0.82]
  Serotype 3: Before 13vPnC dose Year 5 (n=74) | 0.65 [0.56 to 0.76]
  Serotype 3: After 13vPnC dose at Year 5 (n=78) | 1.51 [1.22 to 1.87]
  Serotype 4: After 13vPnC dose at Year 0 (n=79) | 12.81 [9.27 to 17.70]
  Serotype 4: Year 1 (n=74) | 6.00 [4.52 to 7.96]
  Serotype 4: Year 2 (n=75) | 4.63 [3.51 to 6.10]
  Serotype 4: Year 3 (n=77) | 4.12 [3.11 to 5.46]
  Serotype 4: Year 4 (n=76) | 3.82 [2.90 to 5.03]
  Serotype 4: Before 13vPnC dose Year 5 (n=77) | 3.41 [2.61 to 4.46]
  Serotype 4: After 13vPnC dose at Year 5 (n=78) | 24.99 [18.07 to 34.56]
  Serotype 5: After 13vPnC dose at Year 0 (n=82) | 4.21 [3.27 to 5.43]
  Serotype 5: Year 1 (n=75) | 2.43 [2.02 to 2.92]
  Serotype 5: Year 2 (n=78) | 2.05 [1.74 to 2.42]
  Serotype 5: Year 3 (n=79) | 1.86 [1.58 to 2.18]
  Serotype 5: Year 4 (n=78) | 1.84 [1.58 to 2.16]
  Serotype 5: Before 13vPnC dose Year 5 (n=79) | 1.74 [1.47 to 2.08]
  Serotype 5: After 13vPnC dose at Year 5 (n=80) | 5.38 [4.26 to 6.80]
  Serotype 6A: After 13vPnC dose Year 0 (n=82) | 4.32 [3.35 to 5.57]
  Serotype 6A: Year 1 (n=75) | 2.66 [2.15 to 3.27]
  Serotype 6A: Year 2 (n=78) | 2.15 [1.80 to 2.57]
  Serotype 6A: Year 3 (n=79) | 1.96 [1.64 to 2.34]
  Serotype 6A: Year 4 (n=78) | 1.91 [1.62 to 2.26]
  Serotype 6A: Before 13vPnC dose Year 5 (n=79) | 1.74 [1.46 to 2.07]
  Serotype 6A: After 13vPnC dose Year 5 (n=80) | 10.18 [7.50 to 13.82]
  Serotype 6B: After 13vPnC dose Year 0 (n=81) | 5.50 [4.09 to 7.39]
  Serotype 6B: Year 1 (n=74) | 3.24 [2.53 to 4.15]
  Serotype 6B: Year 2 (n=77) | 2.59 [2.13 to 3.16]
  Serotype 6B: Year 3 (n=78) | 2.36 [1.94 to 2.88]
  Serotype 6B: Year 4 (n=77) | 2.20 [1.83 to 2.65]
  Serotype 6B: Before 13vPnC dose Year 5 (n=78) | 1.92 [1.57 to 2.36]
  Serotype 6B: After 13vPnC dose Year 5 (n=79) | 12.82 [9.51 to 17.26]
  Serotype 7F: After 13vPnC dose Year 0 (n=81) | 14.60 [10.96 to 19.46]
  Serotype 7F: Year 1 (n=75) | 6.28 [4.91 to 8.03]
  Serotype 7F: Year 2 (n=77) | 5.03 [3.97 to 6.39]
  Serotype 7F: Year 3 (n=78) | 4.12 [3.30 to 5.15]
  Serotype 7F: Year 4 (n=77) | 3.87 [3.11 to 4.80]
  Serotype 7F: Before 13vPnC dose Year 5 (n=77) | 3.63 [2.92 to 4.50]
  Serotype 7F: After 13vPnC dose Year 5 (n=79) | 11.65 [8.85 to 15.33]
  Serotype 9V: After 13vPnC dose Year 0 (n=80) | 5.81 [4.68 to 7.22]
  Serotype 9V: Year 1 (n=75) | 3.34 [2.80 to 3.98]
  Serotype 9V: Year 2 (n=77) | 2.90 [2.44 to 3.45]
  Serotype 9V: Year 3 (n=77) | 2.60 [2.20 to 3.09]
  Serotype 9V: Year 4 (n=76) | 2.51 [2.14 to 2.94]
  Serotype 9V: Before 13vPnC dose Year 5 (n=77) | 2.24 [1.89 to 2.65]
  Serotype 9V: After 13vPnC dose Year 5 (n=78) | 7.35 [5.92 to 9.12]
  Serotype 14: After 13vPnC dose Year 0 (n=82) | 6.47 [4.43 to 9.46]
  Serotype 14: Year 1 (n=75) | 4.00 [2.86 to 5.59]
  Serotype 14: Year 2 (n=78) | 3.54 [2.61 to 4.82]
  Serotype 14: Year 3 (n=79) | 3.10 [2.28 to 4.22]
  Serotype 14: Year 4 (n=78) | 2.84 [2.10 to 3.83]
  Serotype 14: Before 13vPnC dose Year 5 (n=79) | 2.68 [1.96 to 3.67]
  Serotype 14: After 13vPnC dose Year 5 (n=80) | 6.94 [5.11 to 9.42]
  Serotype 18C: After 13vPnC dose Year 0 (n=82) | 9.86 [7.35 to 13.23]
  Serotype 18C: Year 1 (n=75) | 4.56 [3.54 to 5.87]
  Serotype 18C: Year 2 (n=78) | 3.74 [2.95 to 4.74]
  Serotype 18C: Year 3 (n=79) | 3.11 [2.42 to 4.01]
  Serotype 18C: Year 4 (n=78) | 2.97 [2.38 to 3.71]
  Serotype 18C: Before 13vPnC dose Year 5 (n=79) | 2.77 [2.21 to 3.46]
  Serotype 18C: After 13vPnC dose Year 5 (n=80) | 8.73 [6.64 to 11.48]
  Serotype 19A: After 13vPnC dose Year 0 (n=82) | 5.52 [4.44 to 6.87]
  Serotype 19A: Year 1 (n=75) | 2.69 [2.21 to 3.28]
  Serotype 19A: Year 2 (n=78) | 2.39 [2.00 to 2.85]
  Serotype 19A: Year 3 (n=79) | 2.14 [1.80 to 2.54]
  Serotype 19A: Year 4 (n=78) | 2.06 [1.75 to 2.42]
  Serotype 19A: Before 13vPnC dose Year 5 (n=79) | 1.87 [1.59 to 2.21]
  Serotype 19A: After 13vPnC dose Year 5 (n=80) | 6.00 [4.78 to 7.52]
  Serotype 19F: After 13vPnC dose Year 0 (n=78) | 6.02 [4.68 to 7.75]
  Serotype 19F: Year 1 (n=71) | 3.39 [2.66 to 4.32]
  Serotype 19F: Year 2 (n=72) | 2.74 [2.22 to 3.39]
  Serotype 19F: Year 3 (n=76) | 2.42 [1.97 to 2.98]
  Serotype 19F: Year 4 (n=75) | 2.24 [1.85 to 2.72]
  Serotype 19F: Before 13vPnC dose Year 5 (n=74) | 2.01 [1.59 to 2.55]
  Serotype 19F: After 13vPnC dose Year 5 (n=76) | 18.16 [13.04 to 25.30]
  Serotype 23F: After 13vPnC dose Year 0 (n=80) | 6.65 [5.03 to 8.78]
  Serotype 23F: Year 1 (n=73) | 3.57 [2.90 to 4.40]
  Serotype 23F: Year 2 (n=75) | 3.09 [2.53 to 3.78]
  Serotype 23F: Year 3 (n=77) | 2.93 [2.35 to 3.65]
  Serotype 23F: Year 4 (n=76) | 2.77 [2.23 to 3.46]
  Serotype 23F: Before 13vPnC dose Year 5 (n=77) | 2.48 [2.01 to 3.07]
  Serotype 23F: After 13vPnC dose Year 5 (n=78) | 16.52 [12.29 to 22.22]

21. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Dose 1 (Year 0)
Description: Specific local reactions were prompted for each day,and reported using an electronic diary.Redness and Swelling were scaled as Any(redness present or swelling present);Mild(2.5 to 5.0 centimeters [cm]);Moderate(5.1 to 10.0 cm);Severe (>10 cm). Pain at injection site was scaled as: Any (pain present); Mild (awareness of sign or symptom, but easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating, with inability to do usual activity). Limitation of arm movement was scaled as Any(no limitation of arm movement);Mild(some limitation of arm movement);Moderate (unable to move arm above head but able to move arm above shoulder);Severe (unable to move arm above shoulder). Local reactions were measured only on the participant's arm vaccinated with either 13vPnC or placebo and were not collected at the TIV injection site.
Time Frame: Within 14 days after Dose 1 (Year 0)
Population: Safety population included all participants who had received at least 1 vaccination and did not lack any safety data. Here, n=number of participants with known values.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 551 | 560
percentage of participants
  Redness: Any (n=282,263) | 16.3 | 3.0
  Redness: Mild (n=281,262) | 15.7 | 2.7
  Redness: Moderate (n=265,258) | 4.2 | 0.4
  Redness: Severe (n=262,257) | 0.4 | 0.0
  Swelling: Any (n=288,263) | 18.4 | 3.0
  Swelling: Mild (n=288,263) | 17.0 | 3.0
  Swelling: Moderate (n=263,257) | 5.7 | 0.0
  Swelling: Severe (262,257) | 0.4 | 0.0
  Pain: Any (n=469,321) | 86.8 | 37.1
  Pain: Mild (n=459, 318) | 82.8 | 35.2
  Pain: Moderate (n=324,261) | 39.2 | 4.2
  Pain: Severe (n=267,258) | 4.1 | 0.4
  Limitation of arm movement:Any(317,270) | 35.6 | 8.9
  Limitation of arm movement:Mild(n=310,268) | 32.6 | 8.2
  Limitation of arm movement: Moderate(n=269,259) | 5.2 | 1.2
  Limitation of arm movement:Severe(n=266,258) | 3.4 | 0.8

22. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Dose 2 (Year 0)
Description: as for outcome 21
Time Frame: Within 14 days after Dose 2 (Year 0)
Population: Safety population included all participants who had received at least 1 vaccination and did not lack any safety data. Here,n=number of participants with known values.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 551 | 560
percentage of participants
  Redness: Any (n=238,257) | 1.7 | 12.1
  Redness: Mild (n=238,255) | 1.7 | 10.2
  Redness: Moderate (n=236,248) | 0.0 | 5.6
  Redness: Severe (n=236,242) | 0.0 | 1.2
  Swelling: Any (n=242,265) | 4.5 | 14.7
  Swelling: Mild (n=242,260) | 4.5 | 12.3
  Swelling: Moderate (n=236,249) | 0.4 | 6.4
  Swelling: Severe (236,241) | 0.0 | 0.4
  Pain: Any (n=294,453) | 32.0 | 84.5
  Pain: Mild (n=290, 431) | 30.7 | 82.1
  Pain: Moderate (n=243,319) | 4.5 | 41.1
  Pain: Severe (n=236,248) | 0.0 | 4.8
  Limitation of arm movement:Any(248,318) | 9.3 | 42.5
  Limitation of arm movement:Mild(n=248,316) | 9.3 | 41.1
  Limitation of arm movement: Moderate(n=236,248) | 0.4 | 5.2
  Limitation of arm movement:Severe(n=236,244) | 0.0 | 2.9

23. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After 13vPnC (Year 5)
Description: Specific local reactions were prompted for each day,and reported using an electronic diary.Redness and Swelling were scaled as Any(redness present or swelling present);Mild(2.5 to 5.0 centimeters [cm]);Moderate(5.1 to 10.0 cm);Severe (>10 cm). Pain at injection site was scaled as: Any (pain present); Mild (awareness of sign or symptom, but easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating, with inability to do usual activity). Limitation of arm movement was scaled as Any(no limitation of arm movement);Mild(some limitation of arm movement);Moderate (unable to move arm above head but able to move arm above shoulder);Severe (unable to move arm above shoulder).
Time Frame: Within 14 days after 13vPnC (Year 5)
Population: The safety population at Year 5 included participants who received both (Year 0 and Year 5) 13vPnC and had some safety results at Year 5. Here, n=number of participants with known values.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 364 | 363
percentage of participants
  Redness: Any (n=216,215) | 15.7 | 20.9
  Redness: Mild (n=215,212) | 14.0 | 17.5
  Redness: Moderate (n=210,211) | 7.1 | 12.3
  Redness: Severe (n=205,202) | 1.5 | 0.5
  Swelling: Any (n=224,216) | 18.8 | 18.1
  Swelling: Mild (n=223,214) | 17.5 | 15.9
  Swelling: Moderate (n=211,208) | 7.1 | 9.6
  Swelling: Severe (205,203) | 0.0 | 1.0
  Pain: Any (n=313,306) | 79.2 | 79.4
  Pain: Mild (n=297, 299) | 76.4 | 74.9
  Pain: Moderate (n=248,235) | 32.7 | 34.9
  Pain: Severe (n=206,205) | 4.4 | 3.4
  Limitation of arm movement:Any(233,224) | 23.2 | 26.3
  Limitation of arm movement:Mild(n=233,219) | 22.3 | 22.8
  Limitation of arm movement: Moderate(n=208,206) | 2.9 | 3.9
  Limitation of arm movement:Severe(n=206,206) | 1.9 | 3.4

24. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Dose 1 (Year 0)
Description: Percentage of participants who experienced specific systemic events (mild: 38.0 to 38.4 degrees Celsius [C], moderate: 38.5 to 38.9 degrees C, severe: 39.0 to 40.0 degrees C and potentially life threatening greater than [>] 40.0 degrees C), chills, fatigue, headache, vomiting, decreased appetite, rash, new generalized muscle pain, aggravated generalized muscle pain, new generalized joint pain, and aggravated generalized joint pain prompted for each day were reported using an electronic diary.
Time Frame: Within 14 days after Dose 1 (Year 0)
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 551 | 560
percentage of participants
  Fever: >=38 but <38.5 degree C(n=261,259) | 1.5 | 1.2
  Fever: >=38.5 but <39 degree C(n=262,257) | 1.5 | 0.0
  Fever: >=39 but =<40.0 degree C(n=261,257) | 0.4 | 0.0
  Fever:>40.0 degree C (n=261,257) | 0.0 | 0.4
  Fatigue(n=389,359) | 58.1 | 52.4
  Headache(n=399,382) | 65.9 | 56.5
  Chills(n=306,291) | 31.4 | 21.0
  Rash(n=278,264) | 12.6 | 4.9
  Vomiting(n=266,262) | 5.3 | 3.4
  Decreased appetite(n=315,301) | 30.2 | 22.6
  New generalized muscle pain(n=385,326) | 65.5 | 37.7
  Aggravated generalized muscle pain(n=314,294) | 34.7 | 24.1
  New generalized joint pain(n=309,296) | 33.0 | 24.7
  Aggravated generalized joint pain(n=292,284) | 21.2 | 18.0

25. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Dose 2 (Year 0)
Description: Percentage of participants who experienced specific systemic events (absent: 38.0 degrees Celsius [C], mild: 38.0 to 38.4 degrees C, moderate: 38.5 to 38.9 degrees C, severe: 39.0 to 40.0 degrees C and potentially life threatening > 40.0 degrees C), chills, fatigue, headache, vomiting, decreased appetite, rash, new generalized muscle pain, aggravated generalized muscle pain, new generalized joint pain, and aggravated generalized joint pain prompted for each day were reported using an electronic diary.
Time Frame: Within 14 days after Dose 2 (Year 0)
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 551 | 560
percentage of participants
  Fever: >=38 but <38.5 degree C(n=238,241) | 1.3 | 1.2
  Fever: >=38.5 but <39 degree C(n=239,240) | 1.3 | 0.8
  Fever: >=39 but =<40 degree (n=236,240) | 0.4 | 0.4
  Fever: >40.0 degree C(n=237,240) | 0.4 | 0.0
  Fatigue (n=316,338) | 43.7 | 51.8
  Headache (n=334,338) | 48.2 | 50.9
  Chills (n=273,276) | 20.5 | 24.6
  Rash (n=246,252) | 6.1 | 9.5
  Vomiting (n=247,247) | 6.9 | 6.1
  Decreased appetite(n=270,279) | 20.4 | 25.8
  New generalized muscle pain(n=288,350) | 28.5 | 59.1
  Aggravated generalized muscle pain(n=268,305) | 18.7 | 36.7
  New generalized joint pain(n=268,285) | 20.5 | 27.4
  Aggravated generalized joint pain(n=264,282) | 15.5 | 23.8

26. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After 13vPnC (Year 5)
Description: Percentage of participants who experienced specific systemic events (Fever: >= 38.0 degrees Celsius [C], mild: 38.0 to 38.4 degrees C, moderate: 38.5 to 38.9 degrees C, severe: 39.0 to 40.0 degrees C and potentially life threatening > 40.0 degrees C), chills, fatigue, headache, vomiting, decreased appetite, rash, new generalized muscle pain, aggravated generalized muscle pain, new generalized joint pain, and aggravated generalized joint pain prompted for each day were reported using an electronic diary.
Time Frame: Within 14 days after 13vPnC (Year 5)
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 364 | 363
percentage of participants
  Fever: >= 38.0 degrees C (n=206,209) | 2.4 | 5.3
  Fever: >=38 but <38.5 degree C(n=205,206) | 1.0 | 2.4
  Fever: >=38.5 but <39 degree C(n=206,204) | 0.5 | 2.0
  Fever: >=39 but =<40 degree C(n=205,202) | 0.0 | 0.0
  Fever: >40 degree C(n=205,204) | 1.0 | 1.5
  Fatigue(n=263,251) | 43.7 | 45.8
  Headache(n=256,248) | 46.9 | 51.2
  Chills(n=229,217) | 23.1 | 22.1
  Rash(n=209,210) | 7.7 | 13.8
  Vomiting(n=206,207) | 3.4 | 7.2
  Decreased appetite(n=226,227) | 20.4 | 22.0
  New generalized muscle pain(n=266,253) | 47.7 | 51.0
  Aggravated generalized muscle pain(n=241,223) | 29.9 | 27.4
  New generalized joint pain(n=219,219) | 19.2 | 21.9
  Aggravated generalized joint pain(n=218,214) | 17.4 | 18.2

27. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Acute Pain Within 30 Minutes After Dose 1 (Year 0)
Description: Acute pain was not prompted in the electronic diary however were recorded in a specific page of the case report form (CRF). Acute pain at injection site pain occurred within 30 minutes of vaccination and was scaled as: Any (pain present); Mild (easily tolerated); Moderate (discomfort interfering the usual activity); Severe (Incapacitating with inability to do usual activity). Acute pain was measured only on the participant's arm vaccinated with either 13vPnC or placebo and were not collected at the TIV injection site.
Time Frame: Within 30 Minutes After Dose 1 (Year 0)
Population: Safety population included all participants who had received at least 1 vaccination and did not lack any safety data.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 551 | 560
percentage of participants
  Acute pain (Dose 1):Mild | 6.7 | 6.3
  Acute pain (Dose 1):Moderate | 0.0 | 0.0
  Acute pain (Dose 1):Severe | 0.0 | 0.0
  Acute pain (Dose 1): Any | 6.7 | 6.3

28. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Acute Pain Within 30 Minutes After Dose 2 (Year 0)
Description: as for outcome 27
Time Frame: Within 30 Minutes After Dose 2 (Year 0)
Population: Safety population included all participants who had received at least 1 vaccination (Dose 2, year 0) and did not lack any safety data.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 538 | 543
percentage of participants
  Acute pain (Dose 2):Mild | 5.9 | 6.4
  Acute pain (Dose 2):Moderate | 0.0 | 0.0
  Acute pain (Dose 2):Severe | 0.0 | 0.0
  Acute pain (Dose 2):Any | 5.9 | 6.4

29. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Acute Pain Within 30 Minutes After 13vPnC (Year 5)
Description: Acute pain was not prompted in the electronic diary however were recorded in a specific page of the case report form (CRF). Acute pain at injection site pain occurred within 30 minutes of vaccination and was scaled as: Any (pain present); Mild (easily tolerated); Moderate (discomfort interfering the usual activity); Severe (Incapacitating with inability to do usual activity).
Time Frame: Within 30 Minutes After 13vPnC (Year 5)
Population: Safety population at Year 5 included all participants who had received at least 1 vaccination and did not lack any safety data.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 364 | 363
percentage of participants
  Acute pain at injection site:Mild | 3.8 | 4.4
  Acute pain at injection site:Moderate | 0.3 | 0.0
  Acute pain at injection site:Severe | 0.0 | 0.0
  Acute pain at injection site: Any | 4.1 | 4.4

30. Other Pre Specified Outcome: Percentage of Participants With Serious Adverse Events (SAEs) or Non-serious Adverse Events (Non-SAEs)
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Non-serious AEs are AEs excluding SAEs. In Years 1-4, only deaths and withdrawals due to AEs or SAEs were to be recorded in the case report form.
Time Frame: Signing of informed consent up to 194 days after re-vaccination at Year 5
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV/Placebo (Year 0) and 13vPnC (Year 5) | Placebo+TIV/13vPnC (Year 0) and 13vPnC (Year 5)
Number analyzed (Participants) | 551 | 560
percentage of participants
  SAEs at Dose 1 (Year 0) (n=551,560) | 0.7 | 0.9
  SAEs at Dose 2 (Year 0) (n=538,543) | 0.6 | 1.1
  SAEs at 6-month follow-up (Year 0) (n=538,543) | 3.3 | 1.8
  SAEs at Years 1-4(n=536,542) | 1.5 | 0.6
  SAEs at 13vPnC (Year 5)(n=364,363) | 0.5 | 0.6
  SAEs at 6-month follow-up (Year 5)(n=364,363) | 0.5 | 0.5
  non-SAEs at Dose 1 (Year 0)(n=551,560) | 0.5 | 0.8
  non-SAEs at Dose 2 (Year 0)(n=538,543) | 16.2 | 13.2
  non-SAEs at 6-month follow-up (Year 0)(n=538,543) | 11.3 | 10.9
  non-SAEs at Years 1-4(n=536,542) | 0.2 | 0.0
  non-SAEs at 13vPnC (Year 5)(n=364,363) | 4.7 | 3.6
  non-SAEs at 6-month follow-up (Year 5)(n=364,363) | 0.3 | 68.3

ADVERSE EVENTS:
Time Frame: AEs/SAEs recorded: All AEs for 1 month postvaccination. All SAEs and newly diagnosed chronic medical conditions for 6 months postvaccination. Deaths and withdrawals due to S/AE in Years 1-4
Description: SAEs and AEs were grouped by system organ class and summarized. AEs included AEs collected in electronic diary (local,systemic reactions for 13vPnC; systematic assessment) and AEs collected on case report form at each visit (nonsystematic assessment). Participants who received specified dose and had safety data available were evaluable for safety.
Groups:
- 13vPnC+TIV/Placebo: Dose 1 (Year 0): Participants who received 0.5-mL dose of 13vPnC along with 0.5-mL TIV at Year 0 on Day 1 (Dose 1), were assessed for 1 month after Dose 1.
- 13vPnC+TIV/Placebo: Dose 2 (Year 0): Participants who received 0.5-mL Placebo matched to 13vPnC 1 month after Dose 1 (Dose 2), were assessed for 1 month after Dose 2.
- 13vPnC+TIV/Placebo: 6 Month Follow-up (Year 0): Participants who received 0.5-mL dose of 13vPnC along with 0.5-mL TIV at Year 0 on Day 1, then 0.5-mL Placebo matched to 13vPnC 1 month after, were assessed at the 6-month follow-up visit.
- 13vPnC+TIV/Placebo: Years 1-4: Participants who received 0.5-mL dose of 13vPnC along with 0.5-mL TIV at Year 0 on Day 1, then 0.5-mL Placebo matched to 13vPnC 1 month after, were assessed from 6-month follow-up visit at Year 0 to revaccination with 13vPnC given at Year 5.
- 13vPnC+TIV/Placebo: 13vPnC (Year 5): Participants who received 0.5-mL dose of 13vPnC along with 0.5-mL TIV at Year 0 on Day 1, then 0.5-mL Placebo matched to 13vPnC 1 month after, then 0.5 mL dose of 13vPnC 5 years after initial vaccination, were assessed for 1 month after 13vPnC given at Year 5.
- 13vPnC+TIV/Placebo: 6 Month Follow-up (Year 5): Participants who received 0.5-mL dose of 13vPnC along with 0.5-mL TIV at Year 0 on Day 1, then 0.5-mL Placebo matched to 13vPnC 1 month after, then 0.5 mL dose of 13vPnC 5 years after initial vaccination, were assessed at the 6-month follow-up visit.
- Placebo+TIV/13vPnC: Dose 1 (Year 0): Participants who received 0.5-mL Placebo matched to 13vPnC along with 0.5-mL TIV at Year 0 on Day 1 (Dose 1), were assessed for 1 month after Dose 1.
- Placebo+TIV/13vPnC: Dose 2 (Year 0): Participants who received 0.5-mL dose of 13vPnC 1 month after Dose 1 (Dose 2), were assessed for 1 month after Dose 2.
- Placebo+TIV/13vPnC: 6 Month Follow-up (Year 0): Participants who received 0.5-mL Placebo matched to 13vPnC along with 0.5-mL TIV at Year 0 on Day 1, then 0.5-mL dose of 13vPnC 1 month after, were assessed at the 6-month follow-up visit.
- Placebo+TIV/13vPnC: Years 1-4: Participants who received 0.5-mL Placebo matched to 13vPnC along with 0.5-mL TIV at Year 0 on Day 1, then 0.5-mL dose of 13vPnC 1 month after, were assessed from 6-month follow-up visit at Year 0 to revaccination with 13vPnC given at Year 5.
- Placebo+TIV/13vPnC: 13vPnC (Year 5): Participants who received 0.5-mL Placebo matched to 13vPnC along with 0.5-mL TIV at Year 0 on Day 1, then 0.5-mL dose of 13vPnC 1 month after, then 0.5 mL dose of 13vPnC 5 years after initial vaccination, were assessed for 1 month after 13vPnC given at Year 5.
- Placebo+TIV/13vPnC: 6 Month Follow-up (Year 5): Participants who received 0.5-mL Placebo matched to 13vPnC along with 0.5-mL TIV at Year 0 on Day 1, then 0.5-mL dose of 13vPnC 1 month after, then 0.5 mL dose of 13vPnC 5 years after initial vaccination, were assessed at the 6-month follow-up visit.
Arm/Group | 13vPnC+TIV/Placebo: Dose 1 (Year 0) | 13vPnC+TIV/Placebo: Dose 2 (Year 0) | 13vPnC+TIV/Placebo: 6 Month Follow-up (Year 0) | 13vPnC+TIV/Placebo: Years 1-4 | 13vPnC+TIV/Placebo: 13vPnC (Year 5) | 13vPnC+TIV/Placebo: 6 Month Follow-up (Year 5) | Placebo+TIV/13vPnC: Dose 1 (Year 0) | Placebo+TIV/13vPnC: Dose 2 (Year 0) | Placebo+TIV/13vPnC: 6 Month Follow-up (Year 0) | Placebo+TIV/13vPnC: Years 1-4 | Placebo+TIV/13vPnC: 13vPnC (Year 5) | Placebo+TIV/13vPnC: 6 Month Follow-up (Year 5)
Serious Adverse Events (participants affected / at risk) | 4/551 | 3/538 | 18/538 | 8/536 | 2/364 | 2/364 | 5/560 | 6/543 | 10/543 | 3/542 | 2/363 | 3/363
Other Adverse Events (participants affected / at risk) | 420/551 | 248/538 | 26/538 | 1/536 | 256/364 | 1/364 | 326/560 | 388/543 | 29/543 | 0/542 | 248/363 | 0/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC+TIV/Placebo: Dose 1 (Year 0) (N=551) | 13vPnC+TIV/Placebo: Dose 2 (Year 0) (N=538) | 13vPnC+TIV/Placebo: 6 Month Follow-up (Year 0) (N=538) | 13vPnC+TIV/Placebo: Years 1-4 (N=536) | 13vPnC+TIV/Placebo: 13vPnC (Year 5) (N=364) | 13vPnC+TIV/Placebo: 6 Month Follow-up (Year 5) (N=364) | Placebo+TIV/13vPnC: Dose 1 (Year 0) (N=560) | Placebo+TIV/13vPnC: Dose 2 (Year 0) (N=543) | Placebo+TIV/13vPnC: 6 Month Follow-up (Year 0) (N=543) | Placebo+TIV/13vPnC: Years 1-4 (N=542) | Placebo+TIV/13vPnC: 13vPnC (Year 5) (N=363) | Placebo+TIV/13vPnC: 6 Month Follow-up (Year 5) (N=363)
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peridiverticular abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC+TIV/Placebo: Dose 1 (Year 0) (N=551) | 13vPnC+TIV/Placebo: Dose 2 (Year 0) (N=538) | 13vPnC+TIV/Placebo: 6 Month Follow-up (Year 0) (N=538) | 13vPnC+TIV/Placebo: Years 1-4 (N=536) | 13vPnC+TIV/Placebo: 13vPnC (Year 5) (N=364) | 13vPnC+TIV/Placebo: 6 Month Follow-up (Year 5) (N=364) | Placebo+TIV/13vPnC: Dose 1 (Year 0) (N=560) | Placebo+TIV/13vPnC: Dose 2 (Year 0) (N=543) | Placebo+TIV/13vPnC: 6 Month Follow-up (Year 0) (N=543) | Placebo+TIV/13vPnC: Years 1-4 (N=542) | Placebo+TIV/13vPnC: 13vPnC (Year 5) (N=363) | Placebo+TIV/13vPnC: 6 Month Follow-up (Year 5) (N=363)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 4 | 4 | 0 | 0 | 0 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aggravated generalized joint pain: any (General disorders) | 62/292 | 41/264 | 0 | 0 | 38/218 | 0 | 51/284 | 67/282 | 0 | 0 | 39/214 | 0
Aggravated generalized muscle pain: any (General disorders) | 109/314 | 50/268 | 0 | 0 | 72/241 | 0 | 71/294 | 112/305 | 0 | 0 | 61/223 | 0
Any systemic event (General disorders) | 417/484 | 248/381 | 0 | 0 | 221/307 | 0 | 326/430 | 326/425 | 0 | 0 | 218/290 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0
Chills: any (General disorders) | 96/306 | 56/273 | 0 | 0 | 53/229 | 0 | 61/291 | 68/276 | 0 | 0 | 48/217 | 0
Cyst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite: any (General disorders) | 95/315 | 55/270 | 0 | 0 | 46/226 | 0 | 68/301 | 72/279 | 0 | 0 | 50/227 | 0
Fatigue (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0
Fatigue: any (General disorders) | 226/389 | 138/316 | 0 | 0 | 115/263 | 0 | 188/359 | 175/338 | 0 | 0 | 115/251 | 0
Fever: > 40.0 degrees C (General disorders) | 0/261 | 1/237 | 0 | 0 | 2/205 | 0 | 1/257 | 0/240 | 0 | 0 | 3/204 | 0
Fever: 38.0 to 38.5 degrees C (General disorders) | 4/261 | 3/238 | 0 | 0 | 2/205 | 0 | 3/259 | 3/241 | 0 | 0 | 5/206 | 0
Fever: 38.5 to 39.0 degrees C (General disorders) | 4/262 | 3/239 | 0 | 0 | 1/206 | 0 | 0/257 | 2/240 | 0 | 0 | 4/204 | 0
Fever: 39.0 to 40.0 degrees C (General disorders) | 1/261 | 1/236 | 0 | 0 | 0/205 | 0 | 0/257 | 1/240 | 0 | 0 | 0/202 | 0
Headache: any (General disorders) | 263/399 | 161/334 | 0 | 0 | 120/256 | 0 | 216/382 | 172/338 | 0 | 0 | 127/248 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 3 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site movement impairment (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site nodule (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
New joint pain: any (General disorders) | 102/309 | 55/268 | 0 | 0 | 42/219 | 0 | 73/296 | 78/285 | 0 | 0 | 48/219 | 0
New muscle pain: any (General disorders) | 252/385 | 82/288 | 0 | 0 | 127/266 | 0 | 123/326 | 207/350 | 0 | 0 | 129/253 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Rash: any (General disorders) | 35/278 | 15/246 | 0 | 0 | 16/209 | 0 | 13/264 | 24/252 | 0 | 0 | 29/210 | 0
Vessel puncture site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting: any (General disorders) | 14/266 | 17/247 | 0 | 0 | 7/206 | 0 | 9/262 | 15/247 | 0 | 0 | 15/207 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 7 | 4 | 0 | 0 | 0 | 0 | 5 | 3 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 1 | 1 | 0 | 0 | 0 | 4 | 6 | 2 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 7 | 0 | 0 | 7 | 0 | 4 | 5 | 0 | 0 | 5 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 4 | 0 | 0 | 2 | 0 | 8 | 5 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 8 | 2 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 0 | 0 | 0 | 7 | 3 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 4 | 3 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Any local reaction (Skin and subcutaneous tissue disorders) | 420/474 | 105/300 | 0 | 0 | 256/315 | 0 | 128/325 | 388/456 | 0 | 0 | 248/308 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limitation of arm movement: Any (Skin and subcutaneous tissue disorders) | 113/317 | 23/248 | 0 | 0 | 54/233 | 0 | 24/270 | 135/318 | 0 | 0 | 59/224 | 0
Limitation of arm movement: Mild (Skin and subcutaneous tissue disorders) | 101/310 | 23/248 | 0 | 0 | 52/233 | 0 | 22/268 | 130/316 | 0 | 0 | 50/219 | 0
Limitation of arm movement: Moderate (Skin and subcutaneous tissue disorders) | 14/269 | 1/236 | 0 | 0 | 6/208 | 0 | 3/259 | 13/248 | 0 | 0 | 8/206 | 0
Limitation of arm movement: Severe (Skin and subcutaneous tissue disorders) | 9/266 | 0/236 | 0 | 0 | 4/206 | 0 | 2/258 | 7/244 | 0 | 0 | 7/206 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain: Any (Skin and subcutaneous tissue disorders) | 407/469 | 94/294 | 0 | 0 | 248/313 | 0 | 119/321 | 383/453 | 0 | 0 | 243/306 | 0
Pain: Mild (Skin and subcutaneous tissue disorders) | 380/459 | 89/290 | 0 | 0 | 227/297 | 0 | 112/318 | 354/431 | 0 | 0 | 224/299 | 0
Pain: Moderate (Skin and subcutaneous tissue disorders) | 127/324 | 11/243 | 0 | 0 | 81/248 | 0 | 11/261 | 131/319 | 0 | 0 | 82/235 | 0
Pain: Severe (Skin and subcutaneous tissue disorders) | 11/267 | 0/236 | 0 | 0 | 9/206 | 0 | 1/258 | 12/248 | 0 | 0 | 7/205 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Redness: Any (Skin and subcutaneous tissue disorders) | 46/282 | 4/238 | 0 | 0 | 34/216 | 0 | 8/263 | 31/257 | 0 | 0 | 45/215 | 0
Redness: Mild (Skin and subcutaneous tissue disorders) | 44/281 | 4/238 | 0 | 0 | 30/215 | 0 | 7/262 | 26/255 | 0 | 0 | 37/212 | 0
Redness: Moderate (Skin and subcutaneous tissue disorders) | 11/265 | 0/236 | 0 | 0 | 15/210 | 0 | 1/258 | 14/248 | 0 | 0 | 26/211 | 0
Redness: Severe (Skin and subcutaneous tissue disorders) | 1/262 | 0/236 | 0 | 0 | 3/205 | 0 | 0/257 | 3/242 | 0 | 0 | 1/202 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Swelling: Any (Skin and subcutaneous tissue disorders) | 53/288 | 11/242 | 0 | 0 | 42/224 | 0 | 8/263 | 39/265 | 0 | 0 | 39/216 | 0
Swelling: Mild (Skin and subcutaneous tissue disorders) | 49/288 | 11/242 | 0 | 0 | 39/223 | 0 | 8/263 | 32/260 | 0 | 0 | 34/214 | 0
Swelling: Moderate (Skin and subcutaneous tissue disorders) | 15/263 | 1/236 | 0 | 0 | 15/211 | 0 | 0/257 | 16/249 | 0 | 0 | 20/208 | 0
Swelling: Severe (Skin and subcutaneous tissue disorders) | 1/262 | 0/236 | 0 | 0 | 0/205 | 0 | 0/257 | 1/241 | 0 | 0 | 2/203 | 0
Menopause (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin and subcutaneous tissue disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute pain at injection site (Mild) (General disorders) | 37 | 32 | 0 | 0 | 14 | 0 | 35 | 35 | 0 | 0 | 16 | 0
Acute Pain at injection site (Moderate) (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Pain at injection site (Severe) (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Pain at injection site (Any) (General disorders) | 37 | 32 | 0 | 0 | 15 | 0 | 35 | 35 | 0 | 0 | 16 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.